# Immunotherapy in combination with PARP inhibition in advanced cervical cancer patients functionally competent or deficient for the Fanconi Anemia repair pathway

Protocol Number: 2019-JEK-DIA-001 Protocol Version: Version 1.0 Protocol Version Date: 10 Feb 2020

# **Principal Investigator:**

John P. Diaz, MD Miami Cancer Institute, Baptist Health South Florida 8900 N. Kendall Drive, Miami, FL 33176 786-596-2000

Email: JohnPD@baptisthealth.net

# **Sponsor:**

Miami Cancer Institute, Baptist Health South Florida 8900 N. Kendall Drive, Miami, FL 33176

**IND Number:** 151495

# **Study Funding Provided By:**

Florida Department of Health James & Esther King Biomedical Research Program Grant # 9JK03

# **Study Drug Support Provided By:**

Merck & Co, Inc. Merck Investigator Studies Program # 59481

NCT Number: NCT04483544

#### 1.0 TRIAL SUMMARY

| Abbreviated Title | Pembrolizumab and Olaparib in Cervical Cancer Patients |
|---|---|
| Trial Phase | II |
| Clinical Indication | Cervical Cancer |
| Trial Type | Therapeutic |
| Type of control | None |
| Route of administration | Intravenous and Oral |
| Trial Blinding | None |
| Treatment Groups | One |
| Number of trial participants | 48 |
| Estimated enrollment period | 2-3 years |
| Estimated duration of trial | 3-4 years |
| Duration of Participation | Until lack of clinical benefit is demonstrated. |
| Estimated average length of treatment per patient | 6 months |

#### 2.0 TRIAL DESIGN

The study is a non-randomized, open-label phase II clinical trial of the PD-1 inhibitor pembrolizumab, in combination with the PARP inhibitor olaparib, in patients with stage IV, unresectable or recurrent cervical cancer after failure of first-line therapy.

Patients will be treated with standard doses of pembrolizumab, 200 mg intravenously (IV) every 3 weeks [Chung et al., 2019], which is approved for metastatic cervical cancer patients with PDL-1 expression (CPS  $\geq$ 1) and disease progression on or after chemotherapy. They will also receive olaparib 300mg orally (PO) twice daily (BID), which is the FDA approved dose for treatment of BRCA positive ovarian and breast cancers [Barber et al., 2013; Swisher, 2008; Bouwman et al., 2010; Robson et al., 2017]. One cycle is defined as 3 weeks or 21 days, and both drugs will be started on day 1 of cycle 1. Treatment will be continued until progressive disease or unacceptable toxicity. Evaluation for response with imaging (CT or MRI) will be performed every 9 weeks (3 cycles) using Immune Response Evaluation Criteria (iRECIST) [Seymour et al., 2017]. By this set of criteria, progression will need confirmation with a repeat scan at least four weeks later to rule out the rare but occasionally seen pseudo-progression. New lesions are added to the total burden of disease and only by themselves do not represent progression.

Treatment beyond initial investigator-assessed iRECIST-defined progression will be permitted in a case-by-case basis if the treating physician can document that the patient is experiencing clinical benefit and is tolerating study therapy.

Overlapping toxicities to the combination are not expected. However, the first six patients on the study will be evaluated for any grade 4 hematologic or grade 3 or higher non-hematologic toxicity during the first two cycles of treatment. Adjustment of the doses of olaparib to 300 mg PO daily will be made in subsequent patients if grade 4 hematologic toxicities lasting longer than 7 days, neutropenic fevers or grade 3 non-hematologic toxicities lasting longer than 7 days are observed in at least three of the initial

six patients. If intolerable toxicities arise after three or more cycles in patients otherwise experiencing clinical benefit, patients will have the option of continue pembrolizumab as monotherapy. Special attention will be placed on persistent grade 3 or higher anemia, as myelodysplastic syndromes have been described in around 1.5% of patients receiving olaparib in previous trials[Pujade-Lauraine et al., 2017; Robson et al., 2017; Ledermann et al., 2012; Moore et al., 2014]. Hematologic consultation (with bone marrow aspiration as needed) will be requested for patients developing persistent anemia.

Patients will be followed for three (3) years or until time of death. ORR, PFS, and OS will be determined. Correlative studies will determine the functional status of the Fanconi Anemia pathway promoting homologous recombination repair as well as the microbiome composition in responsive and non-responsive patients. In addition, tumor mutation burden, MSI, and PD-L1 expression will be correlated with Fanconi Anemia pathway status and response to therapy.

# 2.1 Trial Design

The study is a non-randomized, open-label, multi-center, phase II clinical trial of the PD-1 inhibitor pembrolizumab, in combination with the PARP inhibitor olaparib, in patients with stage IV, unresectable or recurrent cervical cancer after failure of first-line therapy.

#### 2.2 Trial Schema



#### 2.3 Schedule of Activities

| Trial Period: | Screening<br>Phase | Treatment Cycles <sup>a</sup> | | | | End of<br>Treatm<br>ent | P | ost-Treat | ment | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | epeate<br>8 cyc | | | Safety | Follow | 0 1 |
| Treatment Cycle/Title: | Screening | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Discon | Follow<br>-up | Up<br>Visits <sup>b</sup> | Survival<br>Follow-Up |
| Scheduling Window (Days): | -28 to -1 | | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | At time of Discon ±7 | 30<br>days<br>post<br>discon<br>±7 | Every 8<br>weeks<br>post<br>discon<br>± 7 | Every 12<br>weeks ±7 |
| <b>Administrative Procedures</b> | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | |
| Medical History | X | X | X | X | X | X | X | X | X | | | | |

| Trial Period: | Screening<br>Phase | | | Tre | atme | nt Cy | clesª | | | End of<br>Treatm<br>ent | F | Post-Treat | ment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | o be r | | | | Safety<br>Follow | Follow<br>Up | Survival |
| Treatment Cycle/Title: | Screening | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Discon | -up | Visits <sup>b</sup> | Follow-Up |
| Scheduling Window (Days): | -28 to -1 | | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | ± 3 | At time of Discon ±7 | 30<br>days<br>post<br>discon<br>±7 | Every 8<br>weeks<br>post<br>discon<br>± 7 | Every 12<br>weeks ±7 |
| Prior and Concomitant Medication Review | X | X | X | X | X | X | X | X | X | | | | |
| Trial Treatment Administration | | X | X | X | X | X | X | X | X | | | | |
| Post-study anticancer therapy status | | - 1 | | | | 21 | 21 | | | | X | X | |
| Survival Status | | | | | | | | | | | X | X | X |
| Clinical Procedures/Assessments | | | | | | | | | | | | | |
| Review Adverse Events | | X | X | X | X | X | X | X | X | X | | | |
| Full Physical Examination | X | | | | | | | | | | | | |
| Directed Physical Examination | | X | X | X | X | X | X | X | X | X | | | |
| Vital Signs and Weight | X | X | X | X | X | X | X | X | X | X | | | |
| ECOG Performance Status | X | X | X | X | X | X | X | X | X | X | | | |
| <b>Laboratory Procedures/Assessments:</b> | analysis perf | forme | d by | LOC | AL la | borat | tory | | | | | | |
| Pregnancy Test – Urine or Serum β-HCG | X <sup>c</sup> | | | | | | | | | | | | |
| PT/INR and aPTT | Xa | | | | | | | | | | | | |
| CBC with Differential | Xa | Xb | X | X | X | X | X | X | X | | | | |
| Comprehensive Serum Chemistry<br>Panel | Xª | X <sup>b</sup> | X | X | X | X | X | X | X | | | | |
| Urinalysis | Xa | | | | | | | | | | | | |
| T3, FT4 and TSH | Xa | | | X | | | Xf | | | | | | |
| Efficacy Measurements | | | | | | | | | | | | | |
| Tumor Imaging | X | | | | X | | | | X <sup>d</sup> | X | | | |
| Tumor Biopsies/Archival Tissue Colle | ection/Correl | ative | Studi | ies Bl | ood | | | | | | | | |
| Archival or Newly Obtained Tissue<br>Collection | Xe | | | | | | | | | | | | |
| Correlative Studies Stool Collection | Xe | | | | Xe | | | | | Xe | | | |
| a Must be performed within | 10.1 | C /1 | ~ | 4.4 | | | ٠., | (0 | 1 1 | D 1) | | l . | |

<sup>&</sup>lt;sup>a</sup> Must be performed within 10 days of the first treatment visit (Cycle 1 Day 1).

<sup>&</sup>lt;sup>b</sup> Hematology (CBC with differential) and Creatinine results must be available and reviewed by the Investigator prior to infusion. A spot creatinine result may be used to proceed with treatment, as Chemistry results may not be available.

<sup>&</sup>lt;sup>c</sup> Must be performed within 72 hours of the first treatment visit (Cycle 1 Day 1).

<sup>&</sup>lt;sup>d</sup> Tumor imaging to be done every 9 weeks (within 1 week before every 4<sup>th</sup> cycle) and will only be required every 12 weeks for patients that have been on treatment for more than 1 year.

<sup>&</sup>lt;sup>e</sup>See Protocol Laboratory Manual.

<sup>&</sup>lt;sup>f</sup> Begining with Cycle 9, T3, FT4 and TSH will be performed every 3 cycles/9 weeks.

# 3.0 OBJECTIVE(S), HYPOTHESIS(ES), AND ENDPOINT(S)

# 3.1 Primary Objective(s), Hypothesis(es), and Endpoint(s)

(1) **Objective:** To determine the ORR through the Immune Response Evaluation Criteria in Solid Tumors (iRECIST) [Seymour et al., 2017].

**Hypothesis:** The combination of PD-1 and PARP inhibition will result in an immune overall response for patients with recurrent cervical carcinoma.

**Primary Endpoint:** Immune overall response rate (iORR)

# 3.2 Secondary Objective(s), Hypothesis(es), and Endpoint(s)

(1) **Objective**: To determine PFS and OS, defined as time from treatment initiation to disease progression or death.

**Hypothesis**: The combination of PD-1 and PARP inhibition will result in a progression-free survival advantage for patients with recurrent cervical carcinoma.

**Secondary Endpoint**: Progression-free survival (PFS)

(2) **Objective**: To evaluate safety and tolerability per the Common Terminology Criteria for Adverse Events (CTCAEv5.0) [Common Terminology Criteria for Adverse Events https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/CTCAE\_v5\_Quick\_Reference\_8.5x11.pdf. Accessed September 30, 2018].

**Hypothesis**: Combination of PD-1 and PARP inhibitors is tolerable in patients with recurrent cervical cancer

**Secondary Endpoint**: Toxicities associated with the regimen

(3) **Objective**: To evaluate if baseline tumor deficiencies in the Fanconi Anemia pathway are associated with antitumor responses to the combination as assessed by the FATSI assay, performed on archived paraffin embedded tumor tissues.

**Hypothesis**: Deficiencies in homologous recombination (HR) repair based on the Fanconi Anemia Triple Stain Immunofluorescence (FATSI) assay will predict a higher iORR to the combination of pembrolizumab and olaparib in patients with cervical cancer.

**Secondary Endpoint**: Immune overall response rate (iORR)

(4) **Objective**: To determine duration of response (DoR).

**Hypothesis**: The combination of PD-1 and PARP inhibition will result in a duration of response (DoR), defined as time from documentation of tumor response to disease progression, in this cohort.

**Secondary Endpoint**: Duration of response (DoR)

# 3.3 Exploratory Objective(s)

(1) **Objective:** To determine whether increased baseline TMB, other deficiencies in DNA damage repair mechanisms and PD-L1 expression correlate with FATSI negativity, and if these findings are independently associated with response to therapy.

#### 4.0 BACKGROUND & RATIONALE

Excitement has been generated following the identification of mutations on the BRCA genes as potential predictors of response to PARP inhibitors and recent clinical trials demonstrating antitumor activity with PARP inhibitors in cancer patients with germline BRCA deficiency [Bryant et al., 2005; Farmer et al., 2005; Tutt et al., 2009; Fong et al., 2009; W Audeh et al., 2010]. The rationale behind these observations is that the BRCA genes are involved in homologous recombination (HR), an example of double-strand break repair, and patients with inherited BRCA germline heterozygocity who developed cancer had acquired BRCA homozygous deficiency in their tumors. The resulting genetic instability becomes an advantage for the tumor to perpetuate. Targeting an additional repair pathway, such as base excision repair through PARP inhibition would induce inability for the tumor to survive, an example of a concept commonly called synthetic lethality. The main role of PARP is to detect and initiate an immediate cellular response to metabolic, chemical, or radiation-induced single-strand breaks by signaling the enzymatic machinery in single-strand breaks.

The BRCA genes collaborate with several others in the Fanconi Anemia (FA) HR pathway [Bagby, D'Andrea et al., 2003; Reid et al., 2007; Xia et al., 2007; Smogorzewska et al., 2007; Kim et al., 2011; Vaz et al., 2010; Machida et al., 2006; Meetei et al., 2004; Garcia-Higuera et al., 2000]. Seventeen complementation groups/genes other interactive proteins have been described. Monoubiquitination of FancD2 and FancI by an FA core complex followed by nuclear localization with other DNA damage



response proteins result in the formation of nuclear repair foci, thus foci formation is the focal functional output of this pathway (Fig 1). Based on this, we developed the FATSI Assay, an immunofluorescence based method that detects FancD2/DAPI/Ki67 and permits the observation of FancD2 foci formation (or lack thereof) in the nucleus of proliferating cells in paraffin embedded tumor tissues [Duan et al., 2013]. We also developed a targeted FA sequencing panel to evaluate potential genetic defects resulting in Fanconi Anemia functional deficiency and confirmed the ability of the FATSI test to enrich for patients exhibiting these alterations at the genomic level.

Supported by an NCI R01 and The NCI Cancer Therapy and Evaluation Center Phase II contract we screened >600 patients in a clinical trial for foci formation deficiency [Villalona-Calero et al.,2016]. Functional deficiency was found in 29% of solid tumor patients. We also showed that it is safe to administer the PARP inhibitor veliparib at doses up to 300 mg per day to patients with FA deficient

tumors, and that veliparib can be safely combined with the DNA damaging agent mitomycin C. Activity was seen for the combination in heavily pretreated patients [Villalona-Calero et al., 2016]. Veliparib as a single agent, showed clinical activity in BRCA/RAD51 germline mutated breast cancer, initially identified through FATSI. However, PARP trapping, rather than PARP inhibition, appears to be a better measure of the activity of PARP inhibitors and veliparib has been demonstrated to be a weaker PARP trapping agent compared to agents such as olaparib and niraparib [Murai et al., 2012; Murai et al., 2014].

# 4.1 Background

Pembrolizumab is a potent humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD-1) receptor, thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2). Based on preclinical in vitro data, pembrolizumab has high affinity and potent receptor blocking activity for PD-1. Pembrolizumab has an acceptable preclinical safety profile and is in clinical development as an intravenous (IV) immunotherapy for advanced malignancies. Pembrolizumab is indicated for the treatment of patients across a number of indications because of its mechanism of action to bind the PD-1 receptor on the T cell. For more details on specific indications refer to the Investigator brochure.

Investigators should be familiar with the current olaparib (AZD2281) Investigator Brochure (IB).

Olaparib (AZD2281, KU-0059436) is a potent Polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerisation (PARP) inhibitor (PARP-1, -2 and -3) that is being developed as an oral therapy, both as a monotherapy (including maintenance) and for combination with chemotherapy and other anticancer agents.

PARP inhibition is a novel approach to targeting tumors with deficiencies in DNA repair mechanisms. PARP enzymes are essential for repairing DNA single strand breaks (SSBs). Inhibiting PARPs leads to the persistence of SSBs, which are then converted to the more serious DNA double strand breaks (DSBs) during the process of DNA replication. During the process of cell division, DSBs can be efficiently repaired in normal cells by homologous recombination repair (HR). Tumors with HR deficiencies (HRD), such as ovarian cancers in patients with BRCA1/2 mutations, cannot accurately repair the DNA damage, which may become lethal to cells as it accumulates. In such tumor types, olaparib may offer a potentially efficacious and less toxic cancer treatment compared with currently available chemotherapy regimens.

BRCA1 and BRCA2 defective tumors are intrinsically sensitive to PARP inhibitors, both in tumor models in vivo [Rottenberg et al., 2008; Hay et al., 2009] and in the clinic [Fong et al., 2009]. The mechanism of action for olaparib results from the trapping of inactive PARP onto the single-strand breaks preventing their repair [Helleday, 2011; Murai et al 2012]. Persistence of SSBs during DNA replication results in their conversion into the more serious DNA DSBs that would normally be repaired by HR repair. Olaparib has been shown to inhibit selected tumor cell lines in vitro and in xenograft and primary explant models as well as in genetic BRCA knock-out models, either as a stand-alone treatment or in combination with established chemotherapies.

A detailed description of the chemistry, pharmacology, efficacy, and safety of olaparib is provided in the Investigator's Brochure.

# 4.1.1 Pharmaceutical and Therapeutic Background

The importance of intact immune surveillance function in controlling outgrowth of neoplastic transformations has been known for decades (Disis, 2010). Accumulating evidence shows a correlation between tumor-infiltrating lymphocytes in cancer tissue and favorable prognosis in various malignancies. In particular, the presence of CD8+ T-cells and the ratio of CD8+ effector T-cells/FoxP3+ regulatory T-cells (T-regs) correlates with improved prognosis and long-term survival in solid malignancies, such as ovarian, colorectal, and pancreatic cancer; hepatocellular carcinoma; malignant melanoma; and renal cell carcinoma. Tumor-infiltrating lymphocytes can be expanded ex vivo and reinfused, inducing durable objective tumor responses in cancers such as melanoma (Dudley et al., 2005; Hunder et al., 2008).

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated T-cells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD-1 (encoded by the gene *Pdcd1*) is an immunoglobulin (Ig) superfamily member related to cluster of differentiation 28 (CD28) and cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) that has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD-L1 and/or PD-L2) [Greenwald et al., 2005; Okazaki et al., 2001].

The structure of murine PD-1 has been resolved (Zhang et al., 2004). PD-1 and its family members are type I transmembrane glycoproteins containing an Ig-variable–type (IgV-type) domain responsible for ligand binding and a cytoplasmic tail responsible for the binding of signaling molecules. The cytoplasmic tail of PD-1 contains 2 tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif, and an immunoreceptor tyrosine-based switch motif. Following T-cell stimulation, PD-1 recruits the tyrosine phosphatases, SHP-1 and SHP-2, to the immunoreceptor tyrosine-based switch motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3 zeta (CD3ζ), protein kinase C-theta (PKCθ), and zeta-chain-associated protein kinase (ZAP70), which are involved in the CD3 T-cell signaling cascade [Okazaki et al., 2001; Chemnitz et al., 2004; Sheppard et al., 2004; and Riley, 2009]. The mechanism by which PD-1 down-modulates T-cell responses is similar to, but distinct from, that of CTLA-4, because both molecules regulate an overlapping set of signaling proteins [Parry et al., 2005; Francisco, 2010]. As a consequence, the PD-1/PD-L1 pathway is an attractive target for therapeutic intervention in cervical cancer.

On June 12, 2018, the FDA approved pembrolizumab for patients with recurrent or metastatic cervical cancer with disease progression on or after chemotherapy whose tumors express PD-L1 (CPS  $\geq$ 1) as determined by an FDA-approved test. The accelerated approval was based on the results of KEYNOTE 158 (NCT02628067). Pembrolizumab was investigated in 98 patients with recurrent or metastatic cervical cancer enrolled in a single cohort of a multicenter, non-randomized, open-label, multi-cohort trial. Patients were treated with pembrolizumab intravenously at a dose of 200 mg every 3 weeks until unacceptable toxicity or documented disease progression [Chung, 2019].

Among the 98 patients, 82 (83.7%) patients had tumors that expressed PD-L1 with a CPS ≥1 PD-L1 status was determined using the PD-L1 IHC 22C3 pharmDx Kit. The major efficacy outcomes were objective response rate (ORR) according to RECIST 1.1 as assessed by blinded independent central review, and response duration. With a median follow-up time of 10.2 months, the ORR was 12.2%

(95% CI: 6.5 to 20.4%), including three complete responses and nine partial responses. All 12 responses were in patients with PDL-1 positive tumors, for an overall response rate of 14.6% (95% CI, 7.8 to 24.2%). The estimated median response duration was not reached (range  $\geq$ 3.7 to  $\geq$  18.6+ months). Treatment related grade 3 to 4 adverse events (diarrhea, asthenia, pyrexia, arthralgias and increase in AST) occurred in 12.2% of patients.

PARP inhibition has been evaluated in several randomized controlled trials. Olaparib was evaluated in two randomized, placebo-controlled double-blind, multi-center studies in patients with recurrent ovarian cancers who were in response to platinum-based therapy. SOLO-2 evaluated patients with a gBRCAm, who had a response to platinum based therapy. These patients were then randomized to maintenance therapy with olaparib. The patient who received olaparib had a PFS 19.1 months compared to 5.5 months in the control arm [Pujade-Lauraine et al., 2017]. STUDY 19 also evaluated olaparib as maintenance therapy for recurrent ovarian cancer, regardless of BRCA status and also demonstrated a PFS advantage to those women receiving olaparib maintenance [Ledermann et al., 2012]. The POLO trial evaluated olaparib for gBRCAm metastatic pancreatic cancer [Golan et al, 2019]. Maintenance olaparib demonstrated a longer PFS for this cohort of pancreatic cancer patients.

#### 4.1.2 Preclinical and Clinical Trial Data

Refer to the Investigator's Brochure for Preclinical and Clinical data.

# 4.1.3 The Interplay between DNA repair deficiency and Immune Checkpoint inhibition

Le et al. reported a Phase II study evaluating the clinical activity of pembrolizumab, in 41 patients with progressive metastatic carcinoma with or without mismatch-repair deficiency [Le et al., 2015]. The immune-related objective response rate and immune-related progression-free survival rate were 40% (4 of 10 patients) and 78% (7 of 9 patients), respectively, for mismatch repair-deficient colorectal cancers and 0% (0 of 18 patients) and 11% (2 of 18 patients) for mismatch repair-proficient colorectal cancers. The median progression-free survival and overall survival were not reached in the cohort with mismatch repair-deficient colorectal cancer but were 2.2 and 5.0 months, respectively, in the cohort with mismatch repair-proficient colorectal cancer.

Interestingly, patients with mismatch repair-deficient non-colorectal cancer had responses similar to those of patients with mismatch repair-deficient colorectal cancer (immune-related objective response rate, 71% [5 of 7 patients]; immune-related progression-free survival rate, 67% [4 of 6 patients]). Whole-exome sequencing revealed a mean of 1782 somatic mutations per tumor in mismatch repair-deficient tumors, as compared with 73 in mismatch repair-proficient tumors (P=0.007), and high somatic mutation loads were associated with prolonged progression-free survival (P=0.02). Since somatic mutations have the potential to encode "non-self" immunogenic antigens the authors hypothesized that tumors with a large number of somatic mutations due to mismatch-repair defects may be susceptible to immune checkpoint blockade.

Vergote et al. is evaluating the combination of pembrolizumab to traditional carboplatin and paclitaxel followed by olaparib maintanence therapy, KEYLYNK-001, as first line treatment in BRCA-nonmutated patients with advanced epithelial ovarian cancer [Vergote et al., 2019]. Similarly, KEYLYNK-009 is evaluating efficacy of olaparib plus pembrolizumab with chemotherapy plus

pembrolizumab after induction with first-line chemotherapy plus pembrolizumab in triple negative breast cancer (TNBC). The primary hypotheses are that olaparib plus pembrolizumab prolongs progression-free survival (PFS) compared with chemotherapy plus pembrolizumab.

#### 4.2 Rationale

#### 4.2.1 Rationale for the Trial and Selected Population

The overarching hypothesis for this trial is that the combination of pembrolizumab and olaparib in patients with advanced cervical cancer will increase the efficacy of pembrolizumab in this population, and that the increase in efficacy will be more marked in those patients harboring recombination repair deficiencies in their tumors. We also hypothesize that the combination will be safe and tolerable without overlapping toxicities. The mechanism for enhanced response to immunotherapy would be primarily through persistence of DNA damage, leading to a greater mutational load and consequently greater neoantigen presentation, recognition by the immune system and improved effector T-cell function leading to tumor cell death. The FATSI assay will identify those patients in which an innate (both somatic or germline) FA pathway repair deficiency exists.

Forty-eight evaluable patients will be enrolled into this study. Patients must have histologically confirmed cervical cancer that is metastatic, unresectable or recurrent and exhibit ECOG performance status (PS) of less than or equal to 2. Patients will be eligible after failure of standard of care first line therapy. Prior therapy with an immune checkpoint inhibitor (PD-1, PDL-1 or PDL-2) is not allowed. PD-L1 positivity is not required for enrollment or treatment, but all patients will have PDL-1 expression assessed by the FDA approved PD-L1 IHC 22C3 pharmDx Kit (Agilent technologies, Carpinteria, CA; standard at our institution). No prior therapy with a PARP inhibitor is allowed.

#### 4.2.2 Justification for Dose

The planned dose of pembrolizumab for this study is 200 mg every 3 weeks (Q3W). Based on the totality of data generated in the Keytruda development program, 200 mg Q3W is the appropriate dose of pembrolizumab for adults across all indications and regardless of tumor type. As outlined below, this dose is justified by:

- Clinical data from 8 randomized studies demonstrating flat dose- and exposure-efficacy relationships from 2 mg/kg Q3W to 10 mg/kg every 2 weeks (Q2W),
- Clinical data showing meaningful improvement in benefit-risk including overall survival at 200 mg Q3W across multiple indications, and
- Pharmacology data showing full target saturation in both systemic circulation (inferred from pharmacokinetic [PK] data) and tumor (inferred from physiologically-based PK [PBPK] analysis) at 200 mg Q3W

Among the 8 randomized dose-comparison studies, a total of 2262 participants were enrolled with melanoma and non-small cell lung cancer (NSCLC), covering different disease settings (treatment naïve, previously treated, PD-L1 enriched, and all-comers) and different treatment settings (monotherapy and in combination with chemotherapy). Five studies compared 2 mg/kg Q3W versus 10 mg/kg Q2W (KN001 Cohort D, KN002, KN010, and KN021), and 3 studies compared 10 mg/kg Q3W versus 10 mg/kg Q2W (KN001 Cohort B3, KN001 Cohort F2 and KN006).

All of these studies demonstrated flat dose- and exposure-response relationships across the doses studied representing an approximate 5- to 7.5-fold difference in exposure. The 2 mg/kg (or 200 mg fixed-dose) Q3W provided similar responses to the highest doses studied. Subsequently, flat dose-exposure-response relationships were also observed in other tumor types including head and neck cancer, bladder cancer, gastric cancer and classical Hodgkin Lymphoma, confirming 200 mg Q3W as the appropriate dose independent of the tumor type. These findings are consistent with the mechanism of action of pembrolizumab, which acts by interaction with immune cells, and not via direct binding to cancer cells.

Additionally, pharmacology data clearly show target saturation at 200 mg Q3W. First, PK data in KN001 evaluating target-mediated drug disposition (TMDD) conclusively demonstrated saturation of PD-1 in systemic circulation at doses much lower than 200 mg Q3W. Second, a PBPK analysis was conducted to predict tumor PD-1 saturation over a wide range of tumor penetration and PD-1 expression. This evaluation concluded that pembrolizumab at 200 mg Q3W achieves full PD-1 saturation in both blood and tumor.

Finally, population PK analysis of pembrolizumab, which characterized the influence of body weight and other participant covariates on exposure, has shown that the fixed-dosing provides similar control of PK variability as weight based dosing, with considerable overlap in the distribution of exposures from the 200 mg Q3W fixed dose and 2 mg/kg Q3W dose. Supported by these PK characteristics, and given that fixed-dose has advantages of reduced dosing complexity and reduced potential of dosing errors, the 200 mg Q3W fixed-dose was selected for evaluation across all pembrolizumab protocols.

The FDA approved dose for treatment of BRCA positive ovarian and breast cancers [Pujade-Lauraine et al., 2017; Ledermann et al., 2012] of olaparib 300mg orally (PO) twice daily (BID) will be utilized.

The dose of olaparib used in this study is 300 mg twice daily which is the currently approved dose.

One cycle is defined as 3 weeks or 21 days, and both drugs (pembrolizumab and olaparib) will be started on day 1 of cycle 1. Overlapping toxicities to the combination are not expected. However, the first six patients on the study will be evaluated for any grade 4 hematologic or grade 3 or higher non-hematologic toxicity during the first two cycles of treatment. Adjustment of the doses of olaparib to 300 mg PO daily will be made in subsequent patients if grade 4 hematologic toxicities lasting longer than 7 days, neutropenic fevers or grade 3 non-hematologic toxicities lasting longer than 7 days are observed in at least three of the initial six patients. If intolerable toxicities arise after three or more cycles in patients otherwise experiencing clinical benefit, patients will have the option to continue pembrolizumab as monotherapy. Special attention will be placed on persistent grade 3 or higher anemia, as myelodysplastic syndromes have been described in around 1.5% of patients receiving olaparib in previous trials [Pujade-Lauraine, et al., 2017; Ledermann et al., 2012; Moore et al., 2014].

#### 4.2.3 Rationale for Endpoints

# 4.2.3.1 Efficacy Endpoints

The primary clinical endpoint is overall Objective Response Rate by iRECIST criteria (iORR).

Secondary clinical endpoints will include Progression Free Survival (PFS) and Overall Survival (OS) and safety and tolerability per the Common Terminology Criteria for Adverse Events (CTCAEv5.0) (Common Terminology Criteria for Adverse Events https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/CTCAE\_v5\_Quick\_Reference 8.5x11.pdf. Accessed September 30, 2018).

Although cervical cancer is curable in early stages, once it has recurred or metastasized less than 20% of patients survive 5 years (Howlader et al., 2017). Pembrolizumab was recently approved for treatment of PD-L1 positive cervical cancer patients in the second line metastatic setting, with an ORR of only 12.2% in the general population on study (Chung et al., 2019). A proposed model to increase pembrolizumab activity is through increasing tumor mutational load and formation of neoantigens expressed on cancer cells, thereby leading to greater recognition of those tumor cells by the immune system (Rizvi et al., 2015; Snyder et al., 2014; Van Allen et al., 2015). This strategy could be achieved through either enriching treated populations with cancer patients harboring innate (germline or somatic) DNA repair deficiencies, by combining immune checkpoint inhibitors with compounds causing DNA damage, such as platinum and other alkylating agents, or using compounds that directly inhibit DNA repair, such as (PARP) inhibitors.

Olaparib is an oral inhibitor of PARP, causing synthetic lethality in BRCA1/2 deficient tumors and is FDA approved for the treatment of metastatic breast and ovarian cancers harboring germline mutations in the BRCA genes or as maintenance in ovarian cancer patients with tumors experiencing prior sensitivity to platinum agents [Pujade-Lauraine et al., 2017; Robson et al., 2017; Ledermann, et al., 2012].

We expect that the combination of pembrolizumab and olaparib in patients with advanced cervical cancer after failure of chemotherapy will lead to increased efficacy compared to single agents in this population, and that the increase in efficacy will be substantial in those patients harboring homologous recombination repair and other deficiencies in DNA damage repair. We also expect that the combination will be safe and tolerable without significant overlapping toxicities.

# 4.2.3.2 Planned Exploratory Biomarker Research

One of the barriers to the generalized applicability of immunotherapy is the identification of patients who will derive the most benefit from this type of therapy, and better predictive biomarkers are urgently needed.

Correlative endpoints in this study will include determining the functional status of the Fanconi Anemia pathway in promoting homologous recombination repair as well as describing the microbiome composition in responsive and non-responsive patients.

#### Fanconi Anemia pathway analysis

The principal correlative endpoint is to evaluate if baseline tumor deficiencies in the FA pathway are associated with antitumor responses to the combination of pembrolizumab and olaparib, as assessed by the FATSI assay performed on archived paraffin embedded tumor tissues.

Since somatic mutations have the potential to encode "non-self" immunogenic antigens, tumors with a large number of somatic mutations due to mismatch-repair defects are predicted to be susceptible to immune checkpoint blockade. Following this logic, tumors with other types of repair deficiency, such as homologous recombination repair would plausibly have a large number of somatic mutations and would likely be susceptible to immune checkpoint blockade.

The FATSI assay has the ability to differentiate between functionally deficient and functionally competent Fanconi Anemia pathway tumors and therefore, could be used to identify additional patients susceptible to pembrolizumab. We hypothesize that the efficacy of immune checkpoint inhibitors could be increased by combining them with compounds causing DNA damage, or compounds causing inhibition of DNA repair such as (PARP) inhibitors. Thus targeting both HR repair and immune checkpoints will result in a synergistic anti-tumor effect. We expect that patients with pre-existing homologous recombination repair as assessed by FATSI would benefit the most from this combination approach.

The FATSI assay will be performed to assess functional deficiency of the FA pathway, as previously described [Duan et al., 2013; Villalona-Calero et al., 2016] using archived paraffin embedded tumors. We hypothesize that a FATSI negative result, correlated with a higher mutational burden, will be associated with a better response rate. FA deficiency in tumors is not required for enrollment on the trial, thus patients with both FA functionally deficient tumors and patients with FA functionally competent tumors will be receiving treatment. Based on prior screening data in solid tumors [Villalona-Calero et al., 2016], we anticipate that approximatively 30% of patients in this trial will be FA functionally deficient.

FFPE tumor tissue will be cut at 4 microns, placed on positively charged slides and stained with hematoxylin and eosin. Additional sections for immunofluorescence staining will be placed in a 60oC oven for 1 h, cooled, deparaffinized and rehydrated through xylenes and graded ethanol solutions to water in standard fashion. Antigen retrieval will be performed by placing slides in Dako's TRS (pH 6.1) antigen retrieval solution (Dako, Carpenteria, CA) in a calibrated vegetable steamer (Black & Decker). Slides will then be placed on a Dako Autostainer for automated staining. Subsequently, tissue sections will be incubated for 1 hour at room temperature with a primary antibody cocktail of rabbit polyclonal FANC-D2 antibody at a dilution of 1:1000 and a monoclonal anti-Ki67 mouse antibody at a dilution of 1:150. Sections will then be co-incubated for 1 hour at room temperature with a secondary antibody (FITC conjugated to anti-rabbit IgG and Alexafluor 594 donkey anti-mouse) at 1:1000. All rinses will be performed on the autostainer with TBST. The sections will be mounted on glass slides using a 4' 6-diamidino-2-phenylindole (DAPI)—containing embedding medium (Vysis Dapi 1, Abbott Laboratories, Downers Grove, IL). FANCD2 foci positive and negative cell lines (MCF-7 and PD20 cells) will be used as controls. Slides will be analyzed under a Nikon E-400 fluorescence microscope. Ki-67 nuclear positivity of greater than 10% (Ki-67/DAPI) is required to consider a sample evaluable. Evaluation of a total of 300 cells (300 DAPI stained nuclei) with less than one foci positive nucleus per 100 cells is the benchmark to define FA pathway deficiency through FATSI.

Exploratory Correlative Endpoints include determining if increased baseline tumor mutation burden (TMB), MSI, and PD-L1 expression correlate with FATSI negativity, and if these findings are independently associated with response to therapy.

#### 5.0 METHODOLOGY

# **5.1 Study Population**

# Diagnosis/Condition for Entry into the Trial

Patients with metastatic or recurrent histologically confirmed cervical carcinoma who have progressed on or after first line standard of care treatment.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

Each patient should meet all of the inclusion criteria and none of the exclusion criteria for this study in order to be assigned to the study intervention. Under no circumstances, can there be exceptions to this rule. Patients who do not meet the entry requirements are screen failures.

# 5.1.1 Participant Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

- 1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of cervical carcinoma will be enrolled in this study.
- 2. Cervical cancer is a disease of the female genital tract. No male patients will be enrolled.
- 3. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:
  - a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
  - b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
- 4. Participant must have recurrent cervical cancer and have a low potential for cure with radiation therapy or surgery alone and:
  - a. May have received up to 2 prior chemotherapy regimens. Platinum sensitizing agents for radiation therapy are considered a chemotherapy regimen.
- 5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol.
- 6. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
- 7. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

- 8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed prior to the first dose of treatment.
- 9. Patient's life expectancy  $\geq$  16 weeks.
- 10. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment. Before patients can be enrolled, they must have normal laboratory values as outlined in Table 1. Labs must also fall within normal limits prior to infusion.

**Table 1 Adequate Organ Function Laboratory Values** 

| System | Laboratory Value |
|---|---|
| Hematological | |
| Absolute neutrophil count (ANC) | ≥1500/µL |
| Platelets | ≥100 000/µL |
| Hemoglobin | ≥9.0 g/dL or ≥5.6 mmol/L <sup>a</sup> |
| Renal | |
| Creatinine <u>OR</u> Measured or calculated <sup>b</sup> creatinine clearance (GFR can also be used in place of creatinine or CrCl) | ≤1.5 × ULN <u>OR</u><br>≥30 mL/min for participant with creatinine<br>levels >1.5 × institutional ULN |
| Hepatic | |
| Total bilirubin | ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN |
| AST (SGOT) and ALT (SGPT) | $\leq$ 2.5 × ULN ( $\leq$ 5 × ULN for participants with liver metastases) |
| Coagulation | |
| International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) | ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants |
| ALT (SCPT)=alanina aminotransfarasa (sarum alutamic nyruwic transaminasa): AST (SCOT)=asnartata | |

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

<sup>&</sup>lt;sup>a</sup> Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.

<sup>&</sup>lt;sup>b</sup> Creatinine clearance (CrCl) should be calculated per institutional standard.

# 5.1.2 Participant Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

- 1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to the first dose of treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
- 2. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
- 3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
- 4. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to the first dose of treatment.

Note: Participants must have recovered from all AEs due to previous therapies to  $\leq$ Grade 1 or baseline. Participants with  $\leq$ Grade 2 neuropathy may be eligible.

Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.

Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment

- 5. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
- 6. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette–Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
- 7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

- 8. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
- 9. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
- 10. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
- 11. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
- 12. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.

Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers

- 13. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
  - Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
- 14. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients, or patients with a known hypersensitivity to olaparib or any of the excipients of the product.
- 15. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.

- 16. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
- 17. Has an active infection requiring systemic therapy.
- 18. Has a known history of Human Immunodeficiency Virus (HIV) infection.

*Note: No HIV testing is required unless mandated by local health authority.* 

Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV), solid organ, and hematopoietic transplant patients.

19. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.

Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.

Patients with known active hepatitis (i.e. Hepatitis B or C).

- Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible.
- Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
- 20. Has a known history of active TB (Bacillus Tuberculosis).
- 21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that interferes with the requirements of the trial or prohibits obtaining informed consent.

- 22. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
- 23. Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

- 24. Has had an allogenic tissue/solid organ/bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
- 25. Resting ECG and EKG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
- 26. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) V. 5.0 grade 2) caused by previous cancer therapy, excluding alopecia.
- 27. Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
- 28. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
- 29. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable).

#### **5.1.3** Lifestyle Considerations

# 5.1.3.1 Meals and Dietary Restrictions

Participants are prohibited to consume grapefruit juice while on olaparib therapy.

Participants should maintain a normal diet unless modifications are required to manage an AE such as diarrhea, nausea or vomiting.

# 5.1.3.2 Contraception

Pembrolizumab may have adverse effects on a fetus in utero. Refer to Appendix 3 for approved methods of contraception.

# 5.1.4 Pregnancy

If a participant inadvertently becomes pregnant while on treatment with pembrolizumab and/or olaparib, the participant will be immediately discontinued from study intervention(s). The site will contact the participant at least monthly and document the participant's status until the pregnancy has been completed or terminated. The outcome of the pregnancy will be reported to Merck within 2 working days if the outcome is a serious adverse experience (e.g. death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn). The study Investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn to Merck

# 5.1.5 Use in Nursing Women

It is unknown whether pembrolizumab or olaparib is excreted in human milk. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, participants who are breast-feeding are not eligible for enrollment.

# **5.2** Trial Intervention(s)

The intervention(s) to be used in this trial is outlined below in Table 2

**Table 2 Trial Intervention(s)** 

| Drug | Dose/Potency | Dose | Route of | Regimen/Treatment | Use |
|---|---|---|---|---|---|
| | | Frequency | Administration | Period | |
| Pembrolizumab | 200 mg | Q3W | IV infusion | Day 1 of each 3-<br>week cycle | Experimental |
| Olaparib tablet | 300 mg | Twice<br>Daily | Oral | Daily | Experimental |

Trial intervention(s) should begin as close as possible to the date on which intervention is assigned.

# **5.2.1** Timing of Dose Administration

Trial interventions should be administered on Day 1 of each cycle after all procedures/assessments have been completed as detailed on the Trial Flow Chart (Section 6.0). Trial interventions may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons.

All trial interventions will be administered on an outpatient basis.

Pembrolizumab 200 mg will be administered as a 30-minute IV infusion every 3 weeks. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).

The Pharmacy Manual contains specific instructions for the preparation of the pembrolizumab infusion fluid and administration of infusion solution.

Pembrolizumab treatment may continue until 24 months of treatment or 35 doses of pembrolizumab, or disease progression, whichever occurs first.

Olaparib will be initiated on cycle 1 day 1 immediately following the completion of the first dose of pembrolizumab. Cycle 1 day 1 infusion should occur in the morning (AM) in order to receive 2 doses on day 1.

Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water. The tablets should be swallowed whole and not chewed, crushed, dissolved or divided. Olaparib tablets can be taken with or without food. If vomiting occurs shortly after the olaparib tablets

are swallowed, the dose should only be replaced if all of the intact tablets can be seen and counted. Should any patient enrolled on the study miss a scheduled dose for whatever reason (e.g., as a result of forgetting to take the tablets or vomiting), the patient will be allowed to take the scheduled dose up to a maximum of 2 hours after that scheduled dose time. If greater than 2 hours after the scheduled dose time, the missed dose is not to be taken and the patient should take their allotted dose at the next scheduled time.

Patients should be given clear instructions on how and when to take their study treatment. Patients will self-administer olaparib.

Any change from the dosing schedule, dose interruptions, dose reductions, dose discontinuations should be recorded in eCRF

# 5.2.2 Dose Modification and toxicity management <u>for immune-related AEs associated with Olaparib and/or Pembrolizumab</u>

# Olaparib Dose Modification

# **Olaparib Dose Reductions**

In case a dose reduction is necessary, olaparib will be administered as follows:

Table 3a Dose reductions for study treatment to manage adverse events

| Initial Dose | Following re-challenge post interruption: Dose reduction 1 | Dose reduction 2 |
|---|---|---|
| 300 mg twice daily | 250 mg twice daily | 200 mg twice daily |

| Table 3b | Dose reduction for study treatment if patient develops moderate r |
|---|---|
| | impairment |

| Initial Dose | Moderate renal impairment (calculated creatinine clearance by Cockcroft -Gault equation or based on a 24 hour urine test between 31 and 50 ml/min): Dose reduction |
|---|---|
| 300 mg twice daily | 200 mg twice daily |

Table 3c Dose reductions for study treatment if patient has to start taking a strong or moderate CYP3A inhibitor

| <b>Initial Dose</b> | Strong CYP3A inhibitor | Moderate CYP3A inhibitor |
|---------------------|------------------------|--------------------------|
| 300 mg twice daily | 100 mg twice daily | 150 mg twice daily |

For guidance on dose reductions for management of AEs (including renal impairment), refer to section 6.2.

For guidance on dose reductions when concomitant strong or moderate CYP3A inhibitors cannot be avoided see section 6.5.

When dose reduction is necessary patients will take one 150 mg tablet and one 100 mg tablet twice daily or two x 100 mg tablet twice daily (see Section 8.4.6), or one 150 mg tablet twice daily or one 100 mg tablet twice daily (see Section 6.5).

#### Pembrolizumab Dose Modification

AEs associated with pembrolizumab exposure may represent an immunologic etiology. These immune-related AEs (irAEs) may occur shortly after the first dose or several months after the last dose of pembrolizumab treatment and may affect more than on body system simultaneously. Therefore, early recognition and initiation of treatment is critical to reduce complications. Based on existing clinical study data, most irAEs were reversible and could be managed with interruptions of pembrolizumab, administration of corticosteroids and/or other supportive care. For suspected irAEs, ensure adequate evaluation to confirm etiology or exclude other causes. Additional procedures or tests such as bronchoscopy, endoscopy, skin biopsy may be included as part of the evaluation. Dose modification and toxicity management guidelines for irAEs associated with pembrolizumab are provided in Table 4.

# Table 4 Dose modification and toxicity management guidelines for immune-related AEs associated with pembrolizumab

#### General instructions:

- 1. Severe and life-threatening irAEs should be treated with IV corticosteroids followed by oral steroids. Other immunosuppressive treatment should begin if the irAEs are not controlled by corticosteroids.
- 2. Pembrolizumab must be permanently discontinued if the irAE does not resolve or the corticosteroid dose is not ≤10 mg/day within 12 weeks of the last pembrolizumab treatment.
- 3. The corticosteroid taper should begin when the irAE is  $\leq$  Grade 1 and continue at least 4 weeks.
- 4. If pembrolizumab has been withheld, pembrolizumab may resume after the irAE decreased to ≤ Grade 1 after corticosteroid taper.

| irAEs | Toxicity grade (CTCAE V5.0) | Action with pembrolizum ab | Corticosteroid<br>and/or other<br>therapies | Monitoring and follow-up |
|---|---|---|---|---|
| Pneumonitis | Grade 2 Grade 3 or 4, or recurrent Grade 2 | Withhold Permanently discontinue | Administer corticosteroids (initial dose of 1 - 2 mg/kg prednisone or equivalent) followed by taper Add prophylactic antibiotics for opportunistic infections | Monitor participants for signs and symptoms of pneumonitis Evaluate participants with suspected pneumonitis with radiographic imaging and initiate corticosteroid treatment |
| Diarrhea /<br>Colitis | Grade 2 or 3 Grade 4 or recurrent Grade 3 | Withhold Permanently discontinue | Administer corticosteroids (initial dose of 1 - 2 mg/kg prednisone or equivalent) followed by taper | <ul> <li>Monitor participants for signs and symptoms of enterocolitis (ie, diarrhea, abdominal pain, blood or mucus in stool with or without fever) and of bowel perforation (ie, peritoneal signs and ileus)</li> <li>Participants with ≥Grade 2 diarrhea suspecting colitis should consider GI consultation and performing endoscopy to rule out colitis</li> <li>Participants with diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be substituted via IV infusion</li> </ul> |

| AST or ALT<br>elevation or<br>Increased<br>Bilirubin | Grade 2 <sup>a</sup> Grade 3 <sup>b</sup> or 4 <sup>c</sup> | Withhold Permanently discontinue | <ul> <li>Administer corticosteroids (initial dose of 0.5 - 1 mg/kg prednisone or equivalent) followed by taper</li> <li>Administer corticosteroids (initial dose of 1 - 2 mg/kg prednisone or equivalent)</li> </ul> | Monitor with liver function tests (consider weekly or more frequently until liver enzyme value returned to baseline or is stable) |
|---|---|---|---|---|
| Type 1<br>diabetes<br>mellitus<br>(T1DM) or<br>Hyperglycemia | New onset T1DM or Grade 3 or 4 hyperglycemia associated with evidence of β-cell failure | Withhold <sup>d</sup> | • Initiate insulin replacement therapy for participants with T1DM • Administer antihyperglycemic in participants with hyperglycemia | Monitor participants for hyperglycemia or other signs and symptoms of diabetes |
| Hypophysitis | Grade 2 Grade 3 or 4 | Withhold or permanently discontinue d | Administer<br>corticosteroids and<br>initiate hormonal<br>replacements as<br>clinically indicated | Monitor for signs and symptoms of hypophysitis (including hypopituitarism and adrenal insufficiency) |
| Hyperthyroidis<br>m | Grade 2 Grade 3 or 4 | Continue Withhold or permanently discontinue d | Treat with non-<br>selective beta-<br>blockers (eg,<br>propranolol) or<br>thionamides as<br>appropriate | Monitor for signs and symptoms of thyroid disorders |

| Hypothyroidis<br>m | Grade 2, 3, or 4 | Continue | • Initiate thyroid replacement hormones (eg, levothyroxine or liothyronine) per standard of care | Monitor for signs and symptoms of thyroid disorders |
|---|---|---|---|---|
| Nephritis and renal dysfunction: grading according to increased creatinine or acute kidney injury | Grade 2 Grade 3 or 4 | Withhold Permanently discontinue | Administer corticosteroids (prednisone 1 – 2 mg/kg or equivalent) followed by taper | Monitor changes of renal function |
| Myocarditis | Grade 1 or 2 Grade 3 or 4 | Withhold Permanently discontinue | Based on severity<br>of AE administer<br>corticosteroids | Ensure adequate evaluation to confirm etiology and/or exclude other causes |
| All Other immune-related AEs | Intolerable/per sistent Grade 2 Grade 3 Grade 4 or recurrent Grade 3 | Withhold or discontinue based on the event e. Permanently discontinue | Based on severity<br>of AE administer<br>corticosteroids | Ensure adequate evaluation to confirm etiology or exclude other causes |

<sup>&</sup>lt;sup>a</sup> AST/ALT: >3.0 - 5.0 x ULN if baseline normal; >3.0 - 5.0 x baseline, if baseline abnormal; bilirubin:>1.5 - 3.0 x ULN if baseline normal; >1.5 - 3.0 x baseline if baseline abnormal

<sup>&</sup>lt;sup>b</sup> AST/ALT: >5.0 to 20.0 x ULN, if baseline normal; >5.0 - 20.0 x baseline, if baseline abnormal; bilirubin:>3.0 - 10.0 x ULN if baseline normal; >3.0 - 10.0 x baseline if baseline abnormal

- <sup>c</sup> AST/ALT: >20.0 x ULN, if baseline normal; >20.0 x baseline, if baseline abnormal; bilirubin: >10.0 x ULN if baseline normal; >10.0 x baseline if baseline abnormal
- <sup>d</sup> The decision to withhold or permanently discontinue pembrolizumab is at the discretion of the investigator or treating physician. For participants with Grade 3 or 4 immune-related endocrinopathy where withhold of pembrolizumab is required, pembrolizumab may be resumed when AE resolves to  $\leq$  Grade 2 and is controlled with hormonal replacement therapy or achieved metabolic control (in case of T1DM)
- <sup>e</sup> Events that require discontinuation include but are not limited to: Guillain-Barre Syndrome, encephalitis, Stevens-Johnson Syndrome and toxic epidermal necrolysis.

# Dose modification and toxicity management of infusion-reactions related to pembrolizumab

Pembrolizumab may cause severe or life-threatening infusion-reactions including severe hypersensitivity or anaphylaxis. Signs and symptoms usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Dose modification and toxicity management guidelines on pembrolizumab associated infusion reaction are provided in Table 5.

Table 5 Pembrolizumab Infusion Reaction Dose modification and Treatment Guidelines

| NCI CTCAE Grade | Treatment | Premedication at Subsequent Dosing |
|---|---|---|
| Grade 1 | Increase monitoring of vital signs as medically indicated until the | None |
| Mild reaction; infusion | participant is deemed medically stable in the opinion of the investigator. | |
| interruption not indicated; | | |
| intervention not indicated | | |
| Grade 2 | Stop Infusion. | Participant may be premedicated 1.5h |
| Requires therapy or infusion | Additional appropriate medical therapy may include but is not limited to: | ( $\pm$ 30 minutes) prior to infusion of |
| interruption but responds | IV fluids | with: |
| promptly to symptomatic | Antihistamines | Diphenhydramine 50 mg po (or |
| treatment (e.g., antihistamines, | NSAIDs | equivalent dose of antihistamine). |
| NSAIDs, narcotics, IV fluids); | Acetaminophen | Acetaminophen 500-1000 mg po (or |
| prophylactic medications | Narcotics | equivalent dose of analgesic). |
| indicated for ≤24 hrs | Increase monitoring of vital signs as medically indicated until the | |
| | participant is deemed medically stable in the opinion of the investigator. | |
| | If symptoms resolve within 1 hour of stopping drug infusion, the infusion | |
| | may be restarted at 50% of the original infusion rate (e.g. from 100 mL/hr | |
| | to 50 mL/hr). Otherwise dosing will be held until symptoms resolve and | |
| | the participant should be premedicated for the next scheduled dose. | |
| | Participants who develop Grade 2 toxicity despite adequate | |
| | premedication should be permanently discontinued from further | |
| | study drug intervention | |
| Grades 3 or 4 | Stop Infusion. | No subsequent dosing |
| Grade 3: | Additional appropriate medical therapy may include but is not limited to: | |
| Prolonged (i.e., not rapidly | Epinephrine** | |
| responsive to symptomatic | IV fluids | |
| medication and/or brief | Antihistamines | |
| interruption of infusion); | NSAIDs | |
| recurrence of symptoms | Acetaminophen | |
| following initial improvement; | Narcotics | |
| hospitalization indicated for | Oxygen | |
| other clinical sequelae (e.g., | Pressors | |
| renal impairment, pulmonary | Corticosteroids | |
| infiltrates) | Increase monitoring of vital signs as medically indicated until the | |
| Grade 4: | participant is deemed medically stable in the opinion of the investigator. | |
| Life-threatening; pressor or | Hospitalization may be indicated. | |
| ventilatory support indicated | **In cases of anaphylaxis, epinephrine should be used immediately. | |
| | Participant is permanently discontinued from further study drug | |
| | intervention. | |

Appropriate resuscitation equipment should be available at the bedside and a physician readily available during the period of drug administration. For further information, please refer to the Common Terminology Criteria for Adverse Events v5.0 (CTCAE) at http://ctep.cancer.gov

# Other allowed dose interruption for pembrolizumab

Pembrolizumab may be interrupted for situations other than treatment-related AEs such as medical / surgical events or logistical reasons not related to study therapy. Participants should be placed back on study therapy within 3 weeks of the scheduled interruption, unless otherwise discussed with the Sponsor. The reason for interruption should be documented in the patient's study record.

#### 5.2.3 Second Course \*

All participants who stop study treatment with SD or better may be eligible for up to an additional 17 cycles (approximately 1 year) of pembrolizumab treatment if they progress after stopping study treatment from the initial treatment phase. This retreatment is termed the Second Course Phase of this study and is only available if the study remains open and the participant meets the following conditions:

#### **Either**

- Stopped initial treatment with study treatment after attaining an investigator-determined confirmed CR based on RECIST 1.1, and
  - Was treated with at least 8 cycles of study treatment before discontinuing treatment, and
  - o Received at least 2 treatments with pembrolizumab beyond the date when the initial CR was declared

#### OR

• Had SD, PR, or CR and stopped study treatment after completion of 35 administrations (approximately 2 years) of study treatment for reasons other than disease progression or intolerability

#### **AND**

- Experienced an investigator-determined radiographic disease progression by iRECIST 1.1 after stopping initial treatment, and
  - At the time of centrally verified disease progression were found to have received pembrolizumab,
     and
  - o No new anticancer treatment was administered after the last dose of study treatment, and
  - The participant meets all of the safety parameters listed in the inclusion criteria and none of the safety parameters listed in the exclusion criteria, and
  - o The study is ongoing

An objective response or disease progression that occurs during the Second Course Phase for a participant will not be counted as an event for the primary analysis of either endpoint in this study.

\*Note: patients must have measurable disease at the start of protocol treatment to be eligible for this provision.

#### 5.3 Randomization or Treatment Allocation

This is a non-randomized trial.

#### 5.4 Stratification

# 5.5 Concomitant Medications/Vaccinations (allowed & prohibited)

Medications or vaccinations specifically prohibited in the exclusion criteria are not allowed during the ongoing trial. If there is a clinical indication for one of these or other medications or vaccinations specifically prohibited during the trial, discontinuation from trial therapy or vaccination may be required. The final decision on any supportive therapy or vaccination rests with the investigator and/or the participant's primary physician. However, the decision to continue the participant on study intervention requires the mutual agreement of the investigator, the Sponsor, and the participant.

# 5.5.1 Acceptable Concomitant Medications

All treatments that the investigator considers necessary for a participant's welfare may be administered at the discretion of the investigator in keeping with the community standards of medical care. All concomitant medication will be recorded on the case report form (CRF) including all prescription, over-the-counter (OTC), herbal supplements, and IV medications and fluids. If changes occur during the trial period, documentation of drug dosage, frequency, route, and date may also be included on the CRF.

The use of any natural/herbal products or other traditional remedies should be discouraged, but use of these products, as well as any medication or vaccine including over-the-counter or prescription medicines, vitamins, and/or herbal supplements that the patient is receiving at the time of enrolment or receives during the study must be recorded along with:

- Reason for use
- Dates of administration including start and end dates
- Dosage information including dose and frequency

#### Anti-emetics/Anti-diarrheals

From screening Part 2 onwards, should a patient develop nausea, vomiting and / or diarrhea, then these symptoms should be reported as AEs (see section 8.3) and appropriate treatment of the event given.

All concomitant medications received within 28 days prior to the first dose of trial intervention and up to 30 days after the last dose of trial intervention should be recorded. Concomitant medications administered after 30 days after the last dose of trial intervention should be recorded for SAEs and Events of Clinical Interest (ECIs) as defined in Section 7.2.

#### **5.5.2** Prohibited Concomitant Medications

Participants are prohibited from receiving the following therapies during the Screening and Treatment Phase (including retreatment for post-complete response relapse) of this trial:

• Antineoplastic systemic chemotherapy or biological therapy

- Immunotherapy not specified in this protocol
- Chemotherapy not specified in this protocol
- Investigational agents other than pembrolizumab and olaparib
- Radiation therapy

Note: Radiation therapy to a symptomatic solitary lesion or to the brain may be allowed at the investigator's discretion.

- Live vaccines within 30 days prior to the first dose of study treatment and while participating in the study. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
- Systemic glucocorticoids for any purpose other than to modulate symptoms from an event of clinical interest of suspected immunologic etiology. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.

Participants who, in the assessment by the investigator, require the use of any of the aforementioned treatments for clinical management should be removed from the study. All treatments that the Investigator considers necessary for a participant's welfare may be administered at the discretion of the Investigator in keeping with the community standards of medical care.

Medications or vaccinations specifically prohibited in the exclusion criteria are not allowed during the ongoing study. If there is a clinical indication for any medication or vaccination specifically prohibited during the study, discontinuation from study therapy or vaccination may be required. The final decision on any supportive therapy or vaccination rests with the investigator and/or the participant's primary physician. However, the decision to continue the participant on study treatment requires the mutual agreement of the investigator, the Sponsor and the participant. However, the decision to continue the participant on study intervention requires the mutual agreement of the investigator, the Sponsor, and the participant.

Medications that may NOT be administered

**Table 6** Prohibited medications

| Prohibited medication/class of drug: | |
|---|---|
| Anticancer therapy: | Not permitted while the patient is receiving study |
| Chemotherapy | medication |
| Immunotherapy | |
| Hormonal therapy* | |
| Radiotherapy (except palliative) | |
| Biological therapy | |
| Other novel agents | |
| Live virus vaccines | Not permitted while the patient is receiving study |
| Live bacterial vaccines | medication and during the 30 day follow up period. |
| | An increased risk of infection by the administration of live virus and bacterial vaccines has been observed with conventional chemotherapy drugs and the effect with olaparib are unknown. |
| | with conventional chemotherapy drugs and the |

<sup>\*</sup>Hormone Replacement Therapy (HRT) is acceptable

Restricted concomitant medications

 Table 7
 Restricted concomitant medications

| Medication/class of drug: | Usage (including limits for duration permitted and special situations in which it's allowed ): |
|---|---|

 Table 7
 Restricted concomitant medications

| Medication/class of drug: | Usage (including limits for duration permitted and special situations in which it's allowed ): |
|---|---|
| Strong CYP3A inhibitors: itraconazole, telithromycin, clarithromycin, boosted protease inhibitors, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir | Strong or moderate CYP3A inhibitors should not be taken with olaparib. If there is no suitable alternative concomitant medication then the dose of olaparib should be reduced for the period of concomitant administration. The dose reduction of olaparib should be recorded in the CRF with the reason documented as concomitant CYP3A inhibitor use. |
| Moderate CYP3A inhibitors: ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil | <ul> <li>Strong CYP3A inhibitors – reduce the dose of olaparib to 100 mg twice daily for the duration of concomitant therapy with the strong inhibitor and for 5 half lives afterwards.</li> <li>Moderate CYP3A inhibitors - reduce the dose of olaparib to 150 mg twice daily for the duration of concomitant therapy with the moderate inhibitor and for 3 half lives afterwards.</li> <li>After the washout of the inhibitor is complete, the olaparib dose can be reescalated.</li> </ul> |
| Strong inducers: phenobarbital, phenytoin, rifampicin, | Strong or moderate CYP3A inducers should not be taken with olaparib. |
| rifabutin, rifapentine, carbamazepine, nevirapine, enzalutamide and St John's Wort | If the use of any strong or moderate CYP3A inducers are considered necessary for the patient's safety and welfare this could diminish the clinical efficacy of olaparib. |
| Moderate CYP3A inducers: bosentan, efavirenz and modafinil | If a patient requires use of a strong or moderate CYP3A inducer then they must be monitored carefully for any change in efficacy of olaparib. |

 Table 7
 Restricted concomitant medications

| Medication/class of drug: | Usage (including limits for duration permitted and special situations in which it's allowed ): |
|---|---|
| <ul> <li>CYP3A4 substrates: hormonal contraceptive, simvastatin, cisapride, cyclosporine, ergot alkaloids, fentanyl, pimozide, sirolimus, tacrolimus and quetiapine</li> <li>CYP2B6 substrates: bupropion,</li> </ul> | Effect of olaparib on other drugs Based on limited <i>in vitro</i> data, olaparib may increase the exposure to substrates of CYP3A4, OATP1B1, OCT1, OCT2, OAT3, MATE1 and MATE2K. Based on limited <i>in vitro</i> data, olaparib may |
| <ul> <li>efavirenz</li> <li>OATP1B1substrates: bosentan, glibenclamide, repaglinide, statins and valsartan</li> <li>OCT1, MATE1 and MATE2K substrates: metformin</li> <li>OCT2 substrates: serum creatinine</li> <li>OAT3 substrates: furosemide, methotrexate</li> </ul> | reduce the exposure to substrates of 2B6. Caution should be observed if substrates of these isoenzymes or transporter proteins are coadministered. |
| Anticoagulant therapy | Patients who are taking warfarin may participate in this trial; however, it is recommended that international normalized ratio (INR) be monitored carefully at least once per week for the first month, then monthly if the INR is stable. Subcutaneous heparin and low molecular weight heparin are permitted. |
| Palliative radiotherapy | Palliative radiotherapy may be used for the treatment of pain at the site of bony metastases that were present at baseline, provided the investigator does not feel that these are indicative of clinical disease progression during the study period. Study treatment should be discontinued for a minimum of 3 days before a patient undergoes therapeutic palliative radiation treatment. Study treatment should be restarted within 4 weeks as long as any bone marrow toxicity has recovered. |

 Table 7
 Restricted concomitant medications

| Medication/class of drug: | Usage (including limits for duration permitted and special situations in which it's allowed ): |
|---|---|
| Administration of other anti-cancer agents | Patients must not receive any other concurrent anti-cancer therapy, including investigational agents, while on study treatment. Patients may continue the use of bisphosphonates or denosumab for bone disease and corticosteroids for the symptomatic control of brain metastases provided the dose is stable before and during the study and they were started at least 4 weeks prior to beginning study treatment. |

There are no prohibited therapies during the Post-Treatment Follow-up Phase.

# 5.5.3 Rescue Medications & Supportive Care

Participants should receive appropriate supportive care measures as deemed necessary by the treating investigator. Suggested supportive care measures for the management of AEs with potential immunologic etiology are outlined along with the dose modification guidelines in Section 5.2.2 (Table 5). Where appropriate, these guidelines include the use of oral or IV treatment with corticosteroids, as well as additional anti-inflammatory agents if symptoms do not improve with administration of corticosteroids. Note that several courses of steroid tapering may be necessary as symptoms may worsen when the steroid dose is decreased. For each disorder, attempts should be made to rule out other causes such as metastatic disease or bacterial or viral infection, which might require additional supportive care. The treatment guidelines are intended to be applied when the Investigator determines the events to be related to pembrolizumab and/or olaparib.

Note: If after the evaluation of the event, it is determined not to be related to pembrolizumab, the Investigator does not need to follow the treatment guidance. Refer to (Table 5) in Section 5.2.2 for guidelines regarding dose modification and supportive care.

It may be necessary to perform conditional procedures such as bronchoscopy, endoscopy, or skin photography as part of evaluation of the event.

#### 5.6 Participant Discontinuation Criteria

Discontinuation of study intervention does not represent withdrawal from the study.

Participants may discontinue study treatment at any time for any reason or be dropped from the study treatment at the discretion of the investigator should any untoward effect occur. In addition, a participant may be discontinued from study treatment by the investigator or the Sponsor if study treatment is inappropriate, the trial plan is violated, or for administrative and/or other safety reasons. Specific details regarding procedures to be performed at study treatment discontinuation are provided in Section 7.1.4 – Other Procedures.

A participant must be discontinued from study treatment but continue to be monitored in the study for any of the following reasons:

- The participant or participant's legally acceptable representative requests to discontinue study treatment
- Confirmed radiographic disease progression outlined in Section 7.1.2.6
- Any progression or recurrence of any malignancy, or any occurrence of another malignancy that requires active treatment
- Unacceptable adverse experiences as described in Section 5.2.2.
- The participant has a medical condition or personal circumstance which, in the opinion of the investigator and/or sponsor, placed the participant at unnecessary risk from continued administration of study treatment.
- The participant has a confirmed positive serum pregnancy test
- Noncompliance with study treatment or procedure requirements
- Recurrent Grade 2 pneumonitis
- Discontinuation of treatment may be considered for participants who have attained a confirmed complete response (CR) and have been treated for at least 8 cycles (at least 24 weeks), receiving 2 cycles of the combination including 2 doses of pembrolizumab and at least 80% of the planned doses of olaparib beyond the date when the initial CR was declared. These participants may be eligible for second course treatment described in Section 5.2.3.
- The participant is lost to follow-up
- Completion of 35 treatments (approximately 2 years) with pembrolizumab

Note: The number of treatments is calculated starting with the first dose. Participants who stop the combination or pembrolizumab after receiving 35 doses may be eligible for retreatment if they progress after stopping study treatment provided they meet the requirements detailed in Section 5.2.3. Participants may be retreated in the Second Course Phase (Retreatment) for up to an additional 17 cycles (approximately 1 year).

- Administrative reasons
- The End of Treatment and Follow-up visit procedures are listed in Section 8 (Protocol Flow Chart) and Section 10.0.1 (Visit Requirements). After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events will be collected for 90 days after the end of treatment). Subjects who discontinue for reasons other than progressive disease will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent or becoming lost to follow-up. After documented disease progression each subject will be followed by telephone for overall survival until death, withdrawal of consent, or the end of the study, whichever occurs first.
## 5.7 Participant withdrawal From Study

A participant must be withdrawn from the study if the participant or the participant's legally acceptable representative withdraws consent from the study.

If a participant withdraws from the study, they will no longer receive study intervention or be followed at scheduled protocol visits.

Specified details regarding procedures to be performed at the time of withdrawal from the study as well as specific details regarding withdrawal from future biomedical research are outlined in Sections 7.1.4.1 and 7.1.4.2.

## Discontinuation of Study Therapy after CR

Discontinuation of treatment may be considered for subjects who have attained a confirmed CR that have been treated for at least 24 weeks with pembrolizumab or the combination and had at least two treatments with pembrolizumab beyond the date when the initial CR was declared.

## 5.8 Participant Replacement Strategy

We anticipate enrollment of 48 patients for which tumor and toxicity assessments following pembrolizumab/olaparib administration can be made. We will replace patients enrolled for which clinical trial discontinuation was performed prior to any administration of pembrolizumab or those for which pembrolizumab is discontinued due to acute hypersensitivity reactions during the first administration of pembrolizumab. An attempt will be made to assess tumor response in all enrolled patients as specified in the protocol. Patients experiencing clinical deterioration after two doses of pembrolizumab, will be considered treatment failures, will count as tumor progression, and will not be replaced.

## 5.9 Clinical Criteria for Early Trial Termination

Early trial termination will be the result of the criteria specified below:

- 1. Quality or quantity of data recording is inaccurate or incomplete
- 2. Poor adherence to protocol and regulatory requirements
- 3. Incidence or severity of adverse drug reaction in this or other studies indicates a potential health hazard to participants
- 4. Plans to modify or discontinue the development of the study drug

In the event of Merck decision to no longer supply either study drug, adequate notification will be provided so that appropriate adjustments to participant treatment can be made.

#### 6.0 TRIAL ASSESSMENTS AND PROCEDURES

#### **6.1 Trial Procedures**

• Study procedures and their timing are summarized in The Trial Flow Chart - Section 6.0.

- Adherence to the study design requirements, including those specified in the Trial Flow Chart, is essential and required for study conduct.
- The investigator is responsible for ensuring that procedures are conducted by appropriately qualified (by education, training, and experience) staff.
- All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria.
- Additional evaluations/testing may be deemed necessary by the investigator, the Sponsor and/or Merck for reasons related to participant safety. In some cases, such evaluation/testing may be potentially sensitive in nature (eg, HIV, Hepatitis C), and thus local regulations may require that additional informed consent be obtained from the participant. In these cases, such evaluations/testing will be performed in accordance with those regulations.

#### **6.1.1** Administrative and General Procedures

#### **6.1.1.1** Informed Consent

The Investigator must obtain documented consent from each potential participant or each participant's legally acceptable representative prior to participating in a clinical trial. If there are changes to a participant's status during the study (e.g. health requirements) the investigator must ensure appropriate consent is in place.

#### **6.1.1.2** General Informed Consent

Consent must be documented by the participant's dated signature or by the participant's legally acceptable representative's dated signature on a consent form along with the dated signature of the person conducting the consent discussion.

A copy of the signed and dated consent form should be given to the participant before participation in the trial.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the participant must receive the IRB/ERC's approval/favorable opinion in advance of use. The participant or his/her legally acceptable representative should be informed in a timely manner if new information becomes available that may be relevant to the participant's willingness to continue participation in the trial. The communication of this information will be provided and documented via a revised consent form or addendum to the original consent form that captures the participant's dated signature or by the participant's legally acceptable representative's dated signature.

Specifics about a trial and the trial population will be added to the consent form template at the protocol level.

The informed consent will adhere to IRB requirements, applicable laws and regulations and Sponsor requirements.

#### 6.1.1.3 Inclusion/Exclusion Criteria

All inclusion and exclusion criteria will be reviewed by the investigator or qualified designee to ensure that the participant qualifies for the trial.

## **6.1.1.4** Medical History

A medical history will be obtained by the investigator or qualified designee. Medical history will include all active conditions, and any condition diagnosed within the prior 10 years that are considered clinically significant by the Investigator. Details regarding the disease for which the participant has enrolled in this study will be recorded separately and not listed as medical history.

## 6.1.1.5 Prior and Concomitant Medications Review

#### 6.1.1.5.1 Prior Medications

The investigator or qualified designee will review prior medication use, including any protocol-specified washout requirement, and record prior medication taken by the participant within 28 days before starting the trial. Treatment for the disease for which the participant has enrolled in this study will be recorded separately and not listed as a prior medication.

#### **6.1.1.5.2** Concomitant Medications

The investigator or qualified designee will record medication, if any, taken by the participant during the trial. In addition, new medication started during the Second Course should be recorded. All medications related to reportable SAEs and ECIs should be recorded as defined in Section 7.2.

#### 6.1.1.6 Disease Details and Treatments

## 6.1.1.6.1 Disease Details

The investigator or qualified designee will obtain prior and current details regarding disease status.

#### 6.1.1.6.2 Prior Treatment Details

The investigator or qualified designee will review all prior cancer treatments including systemic treatments, radiation and surgeries.

# 6.1.1.6.3 Subsequent Anti-Cancer Therapy Status

The investigator or qualified designee will review all new anti-neoplastic therapy initiated after the last dose of trial treatment. If a participant initiates a new anti-cancer therapy within 30 days after the last dose of trial treatment, the 30-day Safety Follow-up visit must occur before the first dose of the new therapy. Once new anti-cancer therapy has been initiated, the participant will move into survival follow-up.

## **6.1.1.7** Assignment of Screening Number

## **6.1.1.8** Assignment of Randomization Number

Not applicable.

## **6.1.1.9** Trial Compliance (Medication/Diet/Activity/Other)

#### 6.1.2 Clinical Procedures/Assessments

# 6.1.2.1 Adverse Event (AE) Monitoring

The investigator or qualified designee will assess each participant to evaluate for potential new or worsening AEs as specified in the Trial Flow Chart and more frequently if clinically indicated. Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to NCI CTCAE Version 5.0 (see Appendix 2). Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment.

Please refer to section 7.2 for detailed information regarding the assessment and recording of AEs.

## 6.1.2.2 Full Physical Exam

The investigator or qualified designee will perform a complete physical exam during the screening period. Clinically significant abnormal findings should be recorded as medical history. A full physical exam should be performed during screening,

## 6.1.2.3 Directed Physical Exam

For cycles that do not require a full physical exam per the Trial Flow Chart, the investigator or qualified designee will perform a directed physical exam as clinically indicated prior to trial treatment administration.

## 6.1.2.4 Vital Signs

The investigator or qualified designee will take vital signs at screening, prior to the administration of each dose of trial treatment and at treatment discontinuation as specified in the Trial Flow Chart (Section 6.0). Vital signs should include temperature, pulse, respiratory rate, weight and blood pressure. Height will be measured at screening only.

## 6.1.2.5 Eastern Cooperative Oncology Group (ECOG) Performance Scale

The investigator or qualified designee will assess ECOG status (see Appendix 1) at screening, prior to the administration of each dose of trial treatment and discontinuation of trial treatment as specified in the Trial Flow Chart.

# 6.1.2.6 Tumor Imaging and Assessment of Disease

Tumor assessments will be performed by computer tomography (CT), PET/CT or Magnetic Resonance Imaging (MRI).

Tumor imaging is strongly preferred to be acquired by computed tomography (CT). For the abdomen and pelvis, contrast-enhanced magnetic resonance imaging (MRI) may be used when CT with iodinated contrast is contraindicated, or when local practice mandates it. MRI is the strongly preferred modality for imaging the brain. The same imaging technique regarding modality, ideally the same scanner, and the use of contrast should be used in a participant throughout the study to optimize the reproducibility of the assessment of existing and new tumor burden and improve the accuracy of the assessment of response or progression based on imaging.

Scans obtained prior to consenting will be allowed, as long as performed within 21 days of study initiation. CT Scans or MRI's will be repeated every 3 cycles (3 weeks cycles); that is before every fourth dose of pembrolizumab in order to assess response to therapy. Tumor imaging will only be required every 12 weeks for patients that have been on treatment for more than 1 year. Immune Response Evaluation Criteria (iRECIST) [36] will be utilized for assessment of response to therapy.

Expedited confirmation of measurable disease based on RECIST 1.1 at Screening should be used to determine participant eligibility. Confirmation that the participant's imaging shows at least 1 lesion that is appropriate for selection as a target lesion per RECIST 1.1 is highly recommended prior to participation allocation.

Participant eligibility will be determined using local assessment (Investigator assessment) based on RECIST 1.1. In addition, images (including via other modalities) that are obtained at an unscheduled time point to determine disease progression, as well as imaging obtained for other reasons, but which demonstrate radiologic progression, should also be used to determine progression.

When the Investigator identifies radiographic progression per RECIST 1.1, efforts should be made to verify radiologic PD. Treatment should continue until PD has been verified. Regardless of whether PD is verified, if the Investigator considers the participant has progressed, but elects to implement iRECIST, the Investigator will assess for confirmation of progression by iRECIST at subsequent time points.

## **6.1.2.6.1** Initial Tumor Imaging

Initial tumor imaging at Screening must be performed within 21 days prior to the date of allocation. The site study team must review screening images to confirm the participant has measurable disease per RECIST 1.1.

The screening images must be submitted to the central imaging vendor for confirmation of measurable disease per RECIST 1.1 for eligibility prior to allocation.

Brain imaging, if performed to document the stability of existing metastases, should be by MRI if possible. If MRI is medically contraindicated, CT with contrast is an acceptable alternative.

## 6.1.2.6.2 Tumor Imaging During the Study

The first on-study imaging assessment should be performed at 9 weeks ( $\pm 7$  days]) from the date of first dose. Subsequent tumor imaging should be performed every 9 weeks ( $\pm 7$  days) or more frequently if clinically indicated. After 52 weeks ( $\pm 7$  days), participants who remain on treatment will have imaging performed every 12weeks ( $\pm 7$  days). Imaging timing should follow calendar days and should not be

adjusted for delays in cycle starts. Imaging should continue to be performed until disease progression is identified by the Investigator.

Objective response should be confirmed by a repeat imaging assessment. Tumor imaging to confirm PR or CR should be performed at least 4 weeks after the first indication of a response is observed. Participants will then return to regular scheduled imaging every 9 weeks, starting with the next scheduled imaging time point. Participants who receive additional imaging for confirmation do not need to undergo the next scheduled tumor imaging if it is less than 4 weeks later; tumor imaging may resume at the subsequent scheduled imaging time point.

Per iRECIST (Section 7.1.2.6.6), disease progression should be confirmed by the site 4 to 8 weeks after first radiologic evidence of PD in clinically stable participants. Participants who have unconfirmed disease progression may continue on treatment at the discretion of the investigator until progression is confirmed by the site provided they have met the conditions detailed in Section 7.1.2.6.6. Participants who receive confirmatory imaging do not need to undergo the next scheduled tumor imaging if it is less than 4 weeks later; tumor imaging may resume at the 1.2.6.6.subsequent scheduled imaging time point, if clinically stable. Participants who have confirmed disease progression by iRECIST, as assessed by the site, will discontinue study treatment. Exceptions are detailed in Section 7.

# 6.1.2.6.3 End of Treatment and Follow-up Tumor Imaging

In participants who discontinue study treatment, tumor imaging should be performed at the time of treatment discontinuation (±4 week window). If previous imaging was obtained within 4 weeks prior to the date of discontinuation, then imaging at treatment discontinuation is not mandatory. In participants who discontinue study treatment due to documented disease progression and the investigator elects not to implement iRECIST, this is the final required tumor imaging.

For participants who discontinue study treatment without documented disease progression, every effort should be made to continue monitoring their disease status by tumor imaging using the same imaging schedule used while on treatment (every 9 weeks in Year 1 or every 12 weeks after Year 1) to monitor disease status until the start of a new anticancer treatment, disease progression, pregnancy, death, withdrawal of consent, or the end of the study, whichever occurs first.

## 6.1.2.6.4 Second Course (Retreatment) Tumor Imaging

Tumor imaging must be performed within 21 days prior to restarting treatment with pembrolizumab. Local reading (Investigator assessment with site radiology reading) will be used to determine eligibility.

The first on-study imaging assessment should be performed at 9 weeks ( $\pm 7$  days) after the restart of treatment. Subsequent tumor imaging should be performed every 9 weeks ( $\pm 7$  days) or more frequently, if clinically indicated.

Per RECIST 1.1 (Section 7.1.2.6.5), if tumor imaging shows initial PD, tumor assessment should be repeated 4 to 8 weeks later in order to confirm PD with the option of continuing treatment while awaiting radiologic confirmation of progression with the option of continuing treatment while awaiting radiological confirmation of progression in clinically stable patients. Participants who obtain confirmatory imaging do not need to undergo scheduled tumor imaging if it is less than 4 weeks later and may wait until the next scheduled imaging time point, if clinically stable.

Imaging should continue to be performed until disease progression, the start of a new anticancer treatment, withdrawal of consent, death, or notification by the Sponsor, whichever occurs first. Disease progression may be confirmed 4 to 8 weeks after the first tumor imaging indicating PD, by the investigator using iRECIST, in clinically stable participants.

In participants who discontinue study treatment, tumor imaging should be performed at the time of treatment discontinuation (±4 week window). If previous imaging was obtained within 4 weeks prior to the date of discontinuation, then imaging at treatment discontinuation is not mandatory. For participants who discontinue study treatment due to documented disease progression, this is the final required tumor imaging.

For participants who discontinue study treatment without documented disease progression, every effort should be made to continue monitoring their disease status by radiologic imaging every 12 weeks (±7 days) until either the start of a new anticancer treatment, disease progression, pregnancy, death, or the end of the study, whichever occurs first.

#### 6.1.2.6.5 RECIST 1.1 Assessment of Disease

RECIST 1.1 will be used as the primary measure for assessment of tumor response, date of disease progression, and as a basis for all protocol guidelines related to disease status (eg, discontinuation of study treatment). Although RECIST 1.1 references a maximum of 5 target lesions in total and 2 per organ, the Sponsor allows a maximum of 10 target lesions in total and 5 per organ, if clinically relevant to enable a broader sampling of tumor burden.

#### 6.1.2.6.6 iRECIST Assessment of Disease

iRECIST is based on RECIST 1.1 but adapted to account for the unique tumor response seen with immunotherapeutic drugs. When clinically stable, participants should not be discontinued until progression is confirmed by the Investigator, working with local radiology, according to the rules below. This allowance to continue treatment despite initial radiologic PD takes into account the observation that some participants can have a transient tumor flare in the first few months after the start of immunotherapy, and then experience subsequent disease response.

A description of the adaptations and iRECIST process is provided in Appendix 4, with additional detail in the iRECIST publication [Seymour et al., 2017]. iRECIST will be used by the Investigator to assess tumor response and progression, and make treatment decisions.

Table 8 Imaging and Treatment after First Radiologic Evidence of Progressive Disease

| | Clinically Stable | | Clinically Unstable | |
|---|---|---|---|---|
| | Imaging | Treatment | Imaging | Treatment |
| First radiologic evidence of PD by RECIST 1.1 | Repeat imaging at 4 to 8 weeks to confirm PD | May continue study treatment at<br>the Investigator's discretion while<br>awaiting confirmatory tumor<br>imaging by site by iRECIST | Repeat imaging at 4 to<br>8 weeks to confirm PD per<br>Investigator's discretion only | Discontinue treatment |
| Repeat tumor imaging<br>confirms PD (iCPD) by<br>iRECIST per Investigator<br>assessment | No additional imaging required | Discontinue treatment (exception is possible upon consultation with Sponsor) | No additional imaging required. | Not applicable |
| Repeat tumor imaging shows iUPD by iRECIST per Investigator assessment | Repeat imaging at 4 to 8 weeks to confirm PD. May occur at next regularly scheduled imaging visit | Continue study treatment at the Investigator's discretion | Repeat imaging at 4 to<br>8 weeks to confirm PD per<br>Investigator's discretion only | Discontinue treatment |
| Repeat tumor imaging shows iSD, iPR, or iCR by iRECIST per Investigator assessment. | Continue regularly scheduled imaging assessments | Continue study treatment at the Investigator's discretion | Continue regularly scheduled imaging assessments. | May restart study treatment if condition has improved and/or clinically stable per Investigator's discretion. Next tumor imaging should occur according to the regular imaging schedule. |

iCPD = iRECIST confirmed progressive disease; iCR = iRECIST complete response; iRECIST = modified Response Evaluation Criteria in Solid Tumors 1.1 for immune-based therapeutics; iSD = iRECIST stable disease; iUPD = iRECIST unconfirmed progressive disease; PD = progressive disease; RECIST 1.1 = Response Evaluation Criteria in Solid Tumors 1.1..

Figure 1: Imaging and Treatment for Clinically Stable Participants after First Radiologic Evidence of PD Assessed by the Investigator



# 6.1.2.7 Tumor Tissue Collection and Correlative Studies Blood Sampling

Formalin fixed paraffin embedded (FFPE) tissue will be obtained from patients participating in the trial. The presence of archival tumor material is part of the criteria for eligibility for this trial.

Stools will be collected prior to the beginning of treatment (within 7 days), after two treatment cycles (prior to the third dose of pembrolizumab) and at the end of treatment.

## **6.1.3** Laboratory Procedures/Assessments

Details regarding specific laboratory procedures/assessments to be performed in this trial are provided below.

Laboratory tests for hematology, chemistry, urinalysis, and others are specified in Table 9.

**Table 9 Laboratory Tests** 

| Hematology | Chemistry | Urinalysis | Other |
|---|---|---|---|
| Hematocrit | Albumin | Blood | Serum β-human chorionic gonadotropin† |
| Hemoglobin | Alkaline phosphatase | Glucose | (β-hCG)† |
| Platelet count | Alanine aminotransferase (ALT) | Protein | PT (INR) |
| WBC (total and differential) | Aspartate aminotransferase (AST) | Specific gravity | aPTT |
| Red Blood Cell Count | Lactate dehydrogenase (LDH) | Microscopic exam (If abnormal) | Total thriiodothyronine (T3) |
| Absolute Neutrophil Count | Carbon Dioxide ‡ | results are noted | Free tyroxine (T4) |
| Absolute Lymphocyte Count | (CO <sub>2</sub> or biocarbonate) | Urine pregnancy test † | Thyroid stimulating hormone (TSH) |
| | Uric Acid | | PK |
| | Calcium | | |
| | Chloride | | Stools for correlative studies |
| | Glucose | | |
| | Phosphorus | | |
| | Potassium | | |
| | Sodium | | |
| | Magnesium | | |
| | Total Bilirubin | | |
| | Direct Bilirubin (If total bilirubin is elevated above the upper limit of normal) | | |
| | Total protein | | |
| | Blood Urea Nitrogen | | |

<sup>†</sup> Perform on women of childbearing potential only. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy test will be required.

<sup>‡</sup> If considered standard of care in your region.

**Table 10 Laboratory safety variables** 

| Haematology/Haemostasis (whole blood) | Clinical Chemistry (serum or plasma) |
|---|---|
| B-Hemoglobin (Hb) | S/P-Creatinine |
| B-Leukocyte count | S/P-Bilirubin, total |
| B-Absolute neutrophil count | S/P-Alkaline phosphatise (ALP) |
| B-Absolute lymphocyte count | S/P-Aspartate transaminase (AST) |
| B-Platelet count | S/P-Alanine transaminase (ALT) |
| B-Mean cell volume (MCV) | S/P-Albumin |
| | S/P-Potassium |
| | S/P-Calcium, total |
| | S/P-Sodium |
| Urinalysis (dipstick) | S/P-Urea or Blood Urea Nitrogen (BUN) |
| U-Hb/Erythrocytes/Blood | S/P-Total Protein |
| U-Protein/Albumin | |
| U-Glucose | |

**NB.** In case a patient shows an AST or ALT  $\ge 3x$ ULN together with total bilirubin  $\ge 2x$ ULN please refer to Appendix E 'Actions required in cases of increases in liver biochemistry and evaluation of Hy's Law', for further instructions.

# 6.1.3.1 Coagulation

- activated partial thromboblastin time {APTT} will be performed at screening and if clinically indicated
- international normalised ratio {INR} will be performed at screening and if clinically indicated. Patients taking warfarin may participate in this study; however, it is recommended that INR be monitored carefully at least once per week for the first month, then monthly if the INR is stable.

Each coagulation test result will be recorded in CRF.

# 6.1.3.2 Bone marrow or blood cytogenetic samples

Bone marrow or blood cytogenetic samples may be collected for patients with prolonged hematological toxicities as defined in Section 8.4.7 per routine medical oncology at Miami Cancer Institute.

Bone marrow analysis should include an aspirate for cellular morphology, cytogenetic analysis and flow cytometry, and a core biopsy for bone marrow cellularity. If it is not possible to conduct cytogenetic analysis or flow cytometry on the bone marrow aspirate, then attempts should be made to carry out the tests on a blood sample. Full reports must be provided by the investigator for documentation on the Patient Safety database. These data are not required to be entered into CRF.

Laboratory tests for screening or entry into the Second Course Phase should be performed within 10 days prior to the first dose of treatment. After Cycle 1, pre-dose laboratory procedures can be conducted up to 72 hours prior to dosing. Results must be reviewed by the investigator or qualified designee and found to be acceptable prior to each dose of trial treatment.

#### **6.1.4** Other Procedures

#### 6.1.4.1 Discontinuation and withdrawal

When a participant discontinues prior to trial completion, all applicable activities scheduled for the final trial visit should be performed at the time of discontinuation. Any adverse events which are present at the time of discontinuation should be followed in accordance with the safety requirements outlined in Section 7.2. - Assessing and Recording Adverse Events. Participants who a) attain a CR or b) complete 24 months of treatment with pembrolizumab may discontinue treatment with the option of restarting treatment if they meet the criteria specified in Section 5.2.3. After discontinuing treatment following assessment of CR, these participants should return to the site for a Safety Follow-up Visit (described in Section 7.1.5.3.1) and then proceed to the Follow-Up Period of the study (described in Section 7.1.5.3.2).

Participants who withdraw prior to completion of the trial should be encouraged to complete all applicable activities scheduled for the final study visit at the time of withdrawal. Any AEs that are present at the time of withdrawal should be followed in accordance with the safety requirements outlined in Section 7.2.

#### 6.1.4.2 Withdrawal from Future Biomedical Research

Participants may withdraw their consent for future biomedical research. Participants may withdraw consent at any time by contacting the investigator. The investigator will inform the Sponsor. It is the responsibility of the investigator to subsequently inform the participant of completion of withdrawal. Any analyses in progress at the time of request for withdrawal or already performed prior to the request for withdrawal being received will continue to be used as part of the overall research study data and results. No new analyses should be generated after the request is received.

In the event that the specimens have been completely anonymized, there will be no link between the participant's personal information and their specimens. In this situation, the request for specimen withdrawal cannot be processed.

#### 6.1.5 Visit Requirements

Visit requirements are outlined in Section 6.0 - Trial Flow Chart. Specific procedure-related details are provided above in Section 7.1 - Trial Procedures.

- 6.1.5.1 Screening
- 6.1.5.1.1 Screening Period
- **6.1.5.2** Treatment Period
- **6.1.5.3** Post-Treatment Visits

## 6.1.5.3.1 Safety Follow-Up Visit

The mandatory Safety Follow-Up Visit should be conducted approximately 30 days after the last dose of study treatment or before the initiation of a new anti-cancer treatment, whichever comes first. All AEs that occur prior to the Safety Follow-Up Visit should be recorded. Participants with an AE of Grade > 1 will be followed until the resolution of the AE to Grade 0-1 or until the beginning of a new anti-cancer therapy, whichever occurs first. SAEs that occur within 90 days of the end of treatment or before initiation of a new anti-cancer treatment should also be followed and recorded. Participants who are eligible for retreatment/crossover with pembrolizumab (as described in Section 5.2.3) may have up to two safety follow-up visits, one after the Initial Treatment Period and one after the Second Course Treatment.

## 6.1.5.3.2 Follow-up Visits

Participants who discontinue study treatment for a reason other than disease progression will move into the Follow-Up Phase and should be assessed every 6 weeks ( $42 \pm 7$  days) by radiologic imaging to monitor disease status. After 1 year, the imaging time point will occur every 9 weeks ( $\pm 7$  days). Every effort should be made to collect information regarding disease status until the start of new anti-cancer therapy, disease progression, death, end of the study or if the participant begins retreatment with pembrolizumab as detailed in Section 5.2.3. Information regarding post-study anti-cancer treatment will be collected if new treatment is initiated.

Participants who are eligible to receive retreatment with pembrolizumab according to the criteria in Section 5.2.3 will move from the follow-up phase to the Second Course Phase when they experience disease progression.

#### 6.1.5.3.3 Survival Follow-up

Participants who experience confirmed disease progression or start a new anticancer therapy, will move into the Survival Follow-Up Phase and should be contacted by telephone every 12 weeks to assess for survival status until death, withdrawal of consent, or the end of the trial, whichever occurs first.

## 6.2 Adverse Events (AEs), Serious Adverse Events (SAEs), and Other Reportable Safety Events

The definitions of an AE or SAE, as well as the method of recording, evaluating, and assessing causality of AE and SAE and the procedures for completing and transmitting AE, SAE, and other reportable safety event reports can be found in Appendix 5.

Adverse events, SAEs, and other reportable safety events will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).

The investigator and any designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE as well as other reportable safety events. Investigators remain responsible for following up AEs, SAEs, and other reportable safety events for outcome.

The investigator, who is a qualified physician, will assess events that meet the definition of an AE or SAE as well as other reportable safety events with respect to seriousness, intensity/toxicity and causality.

#### Olaparib

Any toxicity observed during the course of the study could be managed by interruption of the dose of study treatment or dose reductions. Repeat dose interruptions are allowed as required, for a maximum of 4 weeks on each occasion. If the interruption is any longer, the study team must be informed. Study treatment can be dose reduced to 250 mg twice daily as a first step and to 200 mg twice daily as a second step. If the reduced dose of 200 mg twice daily is not tolerable, no further dose reduction is allowed and study treatment should be discontinued.

Once dose is reduced, escalation is not permitted (except following concomitant treatment with CYP3A4 inhibitors – see Section 6.5

# 6.2.1 Time Period and Frequency for Collecting AE, SAE, and Other Reportable Safety Event Information

All AEs, SAEs, and other reportable safety events that occur after the consent form is signed but before intervention allocation/randomization must be reported by the investigator if the participant is receiving placebo run-in or other run-in treatment, if the event cause the participant to be excluded from the study, or is the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, or a procedure.

- All AEs from the time of intervention allocation/randomization through 30 days following cessation of study intervention must be reported by the investigator.
- All AEs meeting serious criteria, from the time of intervention allocation/randomization through 90 days following cessation of study intervention or 30 days following cessation of study intervention if the participant initiates new anticancer therapy, whichever is earlier, must be reported by the investigator.
- All pregnancies and exposure during breastfeeding, from the time of intervention
  allocation/randomization through 120 days following cessation of study intervention, or 30 days
  following cessation of study intervention if the participant initiates new anticancer therapy must
  be reported by the investigator.
- Additionally, any SAE brought to the attention of an investigator at any time outside of the time
  period specified above must be reported immediately to Merck if the event is considered drugrelated.

Investigators are not obligated to actively seek AEs or SAEs or other reportable safety events in former study participants. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the investigator must promptly notify Merck.

All initial and follow-up AEs, SAEs, and other reportable safety events will be recorded and reported to Merck within the time frames as indicated in Table 11.

Table 11 Reporting Time Periods and Time Frames for Adverse Events and Other Reportable Safety Events

| Type of Event | Reporting Time Period: Consent to Randomization/ Allocation | Reporting Time Period: Randomization/ Allocation through Protocol- specified Follow- up Period | Reporting Time Period: After the Protocol- specified Follow-up Period | Time Frame<br>to Report<br>Event and<br>Follow-up<br>Information<br>to Merck: |
|---|---|---|---|---|
| Serious Adverse Event<br>(SAE) including Cancer<br>and Overdose | Report if: - due to protocol- specified intervention - causes exclusion - participant is receiving placebo run-in or other run- in treatment | Report all | Report if: - drug/vaccine related. (Follow ongoing to outcome) | Within 2<br>business days<br>but no longer<br>than 3<br>calendar days<br>of learning of<br>event |
| Pregnancy/Lactation<br>Exposure | Report if: - due to intervention - causes exclusion | Report all | Previously reported –<br>Follow to<br>completion/termination;<br>report outcome | Within 2<br>business days<br>but no longer<br>than 3<br>calendar days<br>of learning of<br>event |
| Event of Clinical<br>Interest (require<br>regulatory reporting) | Report if: - due to intervention - causes exclusion | Report - potential drug- induced liver injury (DILI) - require regulatory reporting | Not required | Within 2<br>business days<br>but no longer<br>than 3<br>calendar days<br>of learning of<br>event |

## **6.2.1.1** Management of hematological toxicity

# Management of anemia

Table 12 Management of anemia

| Hemoglobin | Action to be taken |
|---|---|
| $\mathbf{Hb} < 10 \ but \ge 8 \ \mathbf{g/dl}$ | First occurrence: |
| (CTCAE Grade 2) | Give appropriate supportive treatment and investigate causality. |
| | Investigator judgement to continue olaparib with supportive treatment (eg transfusion) <i>or</i> interrupt dose for a maximum of 4 weeks. Study treatment can be restarted if Hb has recovered to $> 9g/dl$ . |
| | Subsequent occurrences: |
| | If Hb< 10 $but \ge 9$ g/dl investigator judgement to continue olaparib with supportive treatment (eg transfusion) $or$ dose interrupt (for max of 4 weeks) and upon recovery dose reduction may be considered (to 250 mg twice daily as a first step and to 200 mg twice daily as a second step). |
| | If Hb<9 but $\geq$ 8 g/dl, dose interrupt (for max of 4 weeks) until Hb $\geq$ 9 g/dl and upon recovery dose reduction may be considered (to 250 mg twice daily as a first step and to 200 mg twice daily as a second step). |
| Hb < 8 g/dl<br>(CTCAE Grade 3) | Give appropriate supportive treatment (e.g. transfusion) and investigate causality. |
| , | Interrupt olaparib for a maximum of 4 weeks until improved to $Hb \ge 9$ g/dl. |
| | Upon recovery dose reduce to <b>250 mg twice daily</b> as a first step and to <b>200 mg twice daily</b> as a second step in the case of repeat Hb decrease. |

Common treatable causes of anemia (e.g., iron, vitamin B12 or folate deficiencies and hypothyroidism) should be investigated and appropriately managed. In some cases, management of anemia may require blood transfusions. For cases where patients develop prolonged hematological toxicity (≥2 week interruption/delay in study treatment due to CTC grade 3 or worse anemia and/or development of blood transfusion dependence), refer to guidance later in this section for the management of this.

# Management of neutropenia, leukopenia and thrombocytopenia

Table 13 Management of neutropenia, leukopenia and thrombocytopenia

| Toxicity | Study treatment dose adjustment |
|---|---|
| CTCAE Grade 1-2 | Investigator judgement to continue treatment or if dose interruption, this should be for a maximum of 4 weeks; appropriate supportive treatment and causality investigation |
| CTCAE Grade 3-4 | Dose interruption until recovered to CTCAE gr 1 or better for a maximum of 4 weeks. If repeat CTCAE grade 3-4 occurrence, dose reduce olaparib to <b>250 mg twice daily</b> as a first step and <b>200 mg twice daily</b> as a second step |

Adverse event of neutropenia and leukopenia should be managed as deemed appropriate by the investigator with close follow up and interruption of study drug if CTC grade 3 or worse neutropenia occurs.

Primary prophylaxis with Granulocyte colony-stimulating factor (G-CSF) is not recommended, however, if a patient develops febrile neutropenia, study treatment should be stopped and appropriate management including G-CSF should be given according to local hospital guidelines. Please note that G-CSF should not be used within at least 24 h (7 days for pegylated G-CSF) of the last dose of study treatment unless absolutely necessary.

Platelet transfusions, if indicated, should be done according to local hospital guidelines.

For cases where patients develop prolonged hematological toxicity (≥2 week interruption/delay in study treatment due to CTC grade 3 or worse), refer to guidance later in this section for the management of this.

#### Management of prolonged hematological toxicities while on study treatment

If a patient develops prolonged hematological toxicity such as:

- ≥2 week interruption/delay in study treatment due to CTC grade 3 or worse anaemia and/or development of blood transfusion dependence
- $\geq$ 2 week interruption/delay in study treatment due to CTC grade 3 or worse neutropenia (ANC < 1 x 10<sup>9</sup>/L)
- $\geq$ 2 week interruption/delay in study treatment due to CTC grade 3 or worse thrombocytopenia and/or development of platelet transfusion dependence (Platelets <  $50 \times 10^9$ /L)

Check weekly differential blood counts including reticulocytes and peripheral blood smear. If any blood parameters remain clinically abnormal after 4 weeks of dose interruption, the patient should be referred to hematologist for further investigations. Bone marrow analysis and/or blood cytogenetic analysis should be considered at this stage according to standard hematological practice. Study treatment should be discontinued if blood counts do not recover to CTC gr 1 or better within 4 weeks of dose interruption.

Development of a confirmed myelodysplastic syndrome or other clonal blood disorder should be reported as an SAE and full reports must be provided by the investigator to AstraZeneca Patient Safety. Olaparib treatment should be discontinued if patient's diagnosis of MDS and/or AML is confirmed.

## 6.2.1.2 Management of non-hematological toxicity

Repeat dose interruptions are allowed as required, for a maximum of 4 weeks on each occasion. If the interruption is any longer than this the study monitor must be informed. Where toxicity reoccurs following re-challenge with study treatment, and where further dose interruptions are considered inadequate for management of toxicity, then the patient should be considered for dose reduction or must permanently discontinue study treatment.

Study treatment can be dose reduced to 250 mg twice daily as a first step and to 200 mg twice daily as a second step. Treatment must be interrupted if any NCI-CTCAE grade 3 or 4 adverse event occurs which the investigator considers to be related to administration of study treatment.

## Management of new or worsening pulmonary symptom

If new or worsening pulmonary symptoms (e.g., dyspnea) or radiological abnormalities occur in the absence of a clear diagnosis, an interruption in study treatment dosing is recommended and further diagnostic workup (including a high resolution CT scan) should be performed to exclude pneumonitis.

Following investigation, if no evidence of abnormality is observed on CT imaging and symptoms resolve, then study treatment can be restarted, if deemed appropriate by the investigator. If significant pulmonary abnormalities are identified, these need to be discussed with the Study Physician.

#### Management of nausea and vomiting

Events of nausea and vomiting are known to be associated with olaparib treatment. These events are generally mild to moderate (CTCAE grade 1 or 2) severity, intermittent and manageable on continued treatment. The first onset generally occurs in the first month of treatment for nausea and within the first 6 months of treatment for vomiting. For nausea, the incidence generally plateaus at around 9 months, and for vomiting at around 6 to 7 months.

No routine prophylactic anti-emetic treatment is required at the start of study treatment; however, patients should receive appropriate anti-emetic treatment at the first onset of nausea or vomiting and as required thereafter, in accordance with local treatment practice guidelines. Alternatively, olaparib tablets can be taken with a light meal/snack (i.e. 2 pieces of toast or a couple of biscuits).

As per international guidance on anti-emetic use in cancer patients (ESMO, NCCN), generally a single agent antiemetic should be considered e.g., dopamine receptor antagonist, antihistamines or dexamethasone.

## **Interruptions for intercurrent non-toxicity related events**

Study treatment dose interruption for conditions other than toxicity resolution should be kept as short as possible. If a patient cannot restart study treatment within 4 weeks for resolution of intercurrent conditions not related to disease progression or toxicity, the case should be discussed with AZ study physician.

All dose reductions and interruptions (including any missed doses), and the reasons for the reductions/interruptions are to be recorded in the eCRF.

Study treatment should be stopped at least 3 days prior to planned surgery. After surgery study treatment can be restarted when the wound has healed. No stoppage of study treatment is required for any needle biopsy procedure.

Study treatment should be discontinued for a minimum of 3 days before a patient undergoes radiation treatment. Study treatment should be restarted within 4 weeks as long as any bone marrow toxicity has recovered.

Because the AEs related to olaparib may include asthenia, fatigue and dizziness, patients should be advised to use caution while driving or using machinery if these symptoms occur.

Table 14 Dose reductions for study treatment

| Initial Dose | Following re-challenge post interruption: Dose reduction 1 | Dose reduction 2 |
|---|---|---|
| 300 mg twice daily | 250 mg twice daily | 200 mg twice daily |

## 6.2.1.3 Renal impairment

If subsequent to study entry and while still on study therapy, a patient's estimated CrCl falls below the threshold for study inclusion (≥51 ml/min), retesting should be performed promptly.

A dose reduction is recommended for patients who develop moderate renal impairment (calculated creatinine clearance by Cockcroft-Gault equation or based on a 24-hour urine test of between 31 and 50 ml/min) for any reason during the course of the study: the dose of olaparib should be reduced to 200 mg twice daily.

Because the CrCl determination is only an estimate of renal function, in instances where the CrCl falls to between 31 and 50 mL/min, the investigator should use his or her discretion in determining whether a dose change or discontinuation of therapy is warranted.

Olaparib has not been studied in patients with severe renal impairment (creatinine clearance ≤ 30 ml/min) or end-stage renal disease; if patients develop severe impairment or end stage disease is it recommended that olaparib be discontinued.

# 6.2.2 Method of Detecting AEs, SAEs, and Other Reportable Safety Events

Care will be taken not to introduce bias when detecting AEs and/or SAEs and other reportable safety events. Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about AE occurrence.

## 6.2.3 Follow-up of AE, SAE, and Other Reportable Safety Event Information

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All AEs, SAEs, and other reportable safety events including pregnancy and exposure during breastfeeding, ECIs, cancer, and overdose will be followed until resolution, stabilization, until the event is otherwise explained, or the participant is lost to follow-up. In addition, the investigator will make every attempt to follow all non-serious AEs that occur in randomized participants for outcome. Further information on follow-up procedures is given in Appendix 5.

## **6.2.4** Sponsor Responsibility for Reporting Adverse Events

All AEs will be reported to regulatory authorities, IRB/IECs and investigators in accordance with all applicable country specific regulatory requirements, global laws and regulations.

## 6.2.5 Pregnancy and Exposure During Breastfeeding

Although pregnancy and infant exposure during breastfeeding are not considered AEs, any pregnancy or infant exposure during breastfeeding in a participant (spontaneously reported to the investigator or their designee) that occurs during the study are reportable to Merck.

All reported pregnancies must be followed to the completion/termination of the pregnancy. Pregnancy outcomes of spontaneous abortion, missed abortion, benign hydatidiform mole, blighted ovum, fetal death, intrauterine death, miscarriage, and stillbirth must be reported as serious events (Important Medical Events). If the pregnancy continues to term, the outcome (health of infant) must also be reported.

# **6.2.6** Events of Clinical Interest (ECIs)

Selected non-serious and SAEs are also known as ECIs and must be reported to Merck.

Events of clinical interest for this study include:

- 1. An overdose of pembrolizumab that is not associated with clinical symptoms or abnormal laboratory results. For purposes of this study, an overdose of pembrolizumab will be defined as any dose of 1,000 mg or greater (≥5 times the indicated dose). No specific information is available on the treatment of overdose of pembrolizumab. In the event of overdose, the participant should be observed closely for signs of toxicity. Appropriate supportive treatment should be provided if clinically indicated. If an adverse event(s) is associated with ("results from") the overdose of a Merck product, the adverse event(s) is reported as a serious adverse event, even if no other seriousness criteria are met.
- 2. An elevated AST or ALT lab value that is greater than or equal to 3X the upper limit of normal and an elevated total bilirubin lab value that is greater than or equal to 2X the upper limit of normal and, at the same time, an alkaline phosphatase lab value that is less than 2X the upper limit of normal, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing.\*

\*Note: These criteria are based upon available regulatory guidance documents. The purpose of the criteria is to specify a threshold of abnormal hepatic tests that may require an additional evaluation for an underlying etiology.

There is currently no specific treatment in the event of overdose with olaparib and possible symptoms of overdose are not established.

Olaparib must only be used in accordance with the dosing recommendations in this protocol. Any dose or frequency of dosing that exceeds the dosing regimen specified in this protocol should be reported as an overdose.

Adverse reactions associated with overdose should be treated symptomatically and should be managed appropriately.

#### 7.0 STATISTICAL ANALYSIS PLAN

#### 7.1 Statistical Analysis Plan Summary

# 7.2 Statistical Analysis Plan

Sample size calculation: Single-Stage design will be used for this study [A'Hern, 2001; Fleming, 1982]. The study will require 48 subjects to decide whether the proportion responding (P), is less than or equal to 0.130 or greater than or equal to 0.280. If the number of responses is 10 or more, the hypothesis that P  $\leq$  0.130 is rejected with a target error rate of 0.100 and an actual error rate of 0.087. If the number of responses is nine or less, the hypothesis that P  $\geq$  0.280 is rejected with a target error rate of 0.100 and an actual error rate of 0.099.

<u>Efficacy analyses</u>: The iORR will be defined as the proportion of patients with an "immune" complete response (iCR) or "immune" partial response (iPR). For the primary iORR analysis in all the treated population, patients with an iCR or iPR will be counted as successes and all other patients (including those with missing response information) will be counted as failures. The percentage of iORR with its 95% confidence interval (CI) will be presented.

<u>Progression free survival (PFS)</u> will be defined among all treated patients as the time from first dose of study drug until the first date of either disease progression or death due to any cause. The date of disease progression will be defined as the earliest date of disease progression based on central review. For patients whose disease has not progressed at the time of the analysis, censoring will be performed using the date of the last valid disease assessment. The data will be analyzed by the Kaplan-Meier method. The median PFS time and 95% CI will be recorded.

Overall survival (OS): Median OS will be defined as the time from the beginning of study drug treatment until death due to any cause. For patients who have not died at the time of the analysis, censoring will be performed using the date the patient was last known to be alive. The data will be analyzed by the Kaplan-Meier method. The median OS and 95% CI will be recorded.

<u>Safety analyses:</u> Safety analyses will be presented descriptively. The focus of adverse event (AE) summarization will be on treatment-emergent adverse event (TEAEs). A TEAE is defined as an AE that occurs or worsens in the period extending from the first dose of study drug to 30 days after the last dose of study drug in this study. TEAEs will be summarized and summary tables will be created to show the number of patients reporting TEAEs by severity grade and corresponding percentages. A patient who reports multiple TEAEs within the same Preferred Term (or System Organ Class) is counted only once for that Preferred Term (or System Organ Class) using the worst severity grade. Separate summaries will be prepared for TEAEs classified as severe or life threatening (Grade 3 or higher); study drug-related AEs; AEs leading to treatment interruption, modification, or discontinuation; serious AEs; and death. Dose interruptions, reductions, and relative dose intensity will also be summarized.

All results including efficacy, PFS, OS and safety analysis will also be reported based on race/ethnicity stratification.

<u>FATSI analysis</u> will be conducted in batches. We expect that similar to mismatch repair deficient patients, the immune-related objective response will be at or above 40% in patients with functional FA deficiency (FATSI negative), and less than 10% in patients without either homologous recombination repair

deficiency or mismatch repair deficiency. Based on our prior screening data, we anticipate that close to 30% of patients will be FA functionally deficient.

Total enrollment of 48 patients is planned. We will report the 90% confidence interval estimates of iORR both overall and by FATSI status using the exact method (Clopper Pearson). However, the planned study is small for a well powered comparison given that we expect only 15 FATSI-negative patients. Instead, variation in iORR by FATSI status will be assessed by considering the one-sided 95% lower confidence limit (95%LCL) for the difference. As an example, an observed increase in iORR for FATSI- patients of 30.9%, based on 6 out of 15 FATSI- responders compared with 3 out of 33 FATSI+ responders, provides 95% confidence that the true increase for patients with FA deficient tumors is at least 7.1%, suggesting that further study of pembrolizumab/olaparib in FA deficient cervical cancer patients is warranted.

Kaplan-Meier curves will be used to estimate the distributions of overall survival and immune-related progression-free survival (iPFS). Point estimates and 2-sided 95% confidence intervals will be reported for selected times using Greenwood's variance and the log-log transform method. This will include the 20-week iPFS for purposes of comparison. Based on the panel sequencing results, somatic alterations will be summarized and reported as proportions for genes in FA competent and FA functionally deficient tumors. Confidence intervals will be calculated using the exact method. Additional analyses will be done to establish relationships between treatment and certain baseline characteristics, including deficiencies in the FA pathway, PD-L1 expression, TMB, other deficiencies in DNA damage repair mechanisms. These relationships will be explored primarily through logistic regression or cox proportional hazards regression, depending on the outcome of interest.

For known or predicted deleterious mutations of suspected inheritance trait detected during the trial, the process would be aided by making sure that patients carrying these mutations get referred for genetic counseling and CLIA certified germline analysis. The Miami Cancer Institute has these services readily available.

Stool Microbiome Data Analyses: Centered log-ratio (CLR) transformations will be applied to microbiome data. Log-ratios make the data symmetric and linearly related, and places the data in a log-ratio coordinate space. Thus, we can obtain information about the log-ratio abundances of features relative to other features in the compositional dataset. Zero counts of operational taxonomic units (OTU) will be converted to a probability vector prior to centered log-ratio transformation. Aitchison distance, which is simply the Euclidian distance between samples after CLR transformation, and the distances between samples same as the phylogenetic isometric log-ratio (ILR), will be calculated and used for clustering and ordination. Compositional principal component analysis (PCA) will be applied and biplots will be used to display the relationships between OTUs and the distances between samples.

Differential relative abundance will be based on the CLR values from a modelled probability distribution of the dataset, and the expected values of parametric and non-parametric statistical tests along with effect-size estimates will be reported. This approach reduces the false-positive identification problem to near 0 in real and modelled microbiome datasets with little effect of sensitivity to the negative correlation bias and is observed to be relatively insensitive to change when the data are subset.

Considering possible correlations among metabolites, penalized logistic model will be applied for selecting compositional components, which can predict the status of response to treatment and of treatment

related toxicity. The penalization coefficient  $\lambda$  is selected through leaving-one-out cross-validation.  $\lambda$ , which gives the smallest conditional likelihood deviance, will be used in final prediction.

Penalized survival models will be applied to investigate potential compositional components, which are associated with PFS. Similar to penalized logistic models, penalization hyperparameters will be selected through leaving-one-out cross-validation.

## 8.0 LABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL SUPPLIES

## 8.1 Investigational Product

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of investigational product in accordance with the protocol and any applicable laws and regulations.

Pembrolizumab and olaparib will be provided by Merck as summarized in Table 15.

**Table 15 Product Descriptions** 

| Product Name & Potency | Dosage Form |
|---------------------------------|------------------------|
| Pembrolizumab 100 mg/ 4mL | Solution for Injection |
| Olaparib 100 and 150 mg tablets | Oral |

# 8.2 Packaging and Labeling Information

Supplies will be labeled in accordance with regulatory requirements.

#### 8.3 Clinical Supplies Disclosure

This trial is open-label; therefore, the participant, the trial site personnel, the Sponsor and/or designee are not blinded to treatment. Drug identity (name, strength) is included in the label text; random code/disclosure envelopes or lists are not provided.

## 8.4 Storage and Handling Requirements

Clinical supplies must be stored in a secure, limited-access location under the storage conditions specified on the label.

Receipt and dispensing of trial medication must be recorded by an authorized person at the trial site.

Clinical supplies may not be used for any purpose other than that stated in the protocol.

#### 8.5 Returns and Reconciliation

The Miami Cancer Institute has a dedicated Investigational Drug Service (IDS), including a dedicated IDS Supervisor who leads the coordination of investigational drugs services for clinical research at Miami Cancer Institute (including inventory and receipt as detailed below).

Investigational Drug Services (IDS) Supervisor:

Nicholas Chow, Pharm D, BCOP 8900 N. Kendall Drive Miami, FL 33176 Office: (786) 527-7615

Email: nicholascho@baptisthealth.net

The IDS team provides required pharmacy services for investigational drug studies including oversight of drug storage, handling, preparation, deposition, medication dosing, staff education, and other related activities. All pharmacists involved in the compounding of investigational products are trained on each individual protocol in regards to receipt, preparation, storage, dispensing and administration, product reconciliation and source documentation. Additionally, all pharmacists involved in the compounding aspect are CITI trained and listed on the delegation of authority.

- Disposition and/or destruction of IPs following drug accountability are performed according to specific instructions provided by the sponsor and/or protocol. Disposal and/or destruction of investigational products on-site are performed in accordance with BHM BCH administrative policy
- All products will be disposed of according to regulatory requirements according to institutional policy and in accordance with the Environmental Protection Agency and the State of Florida Department of Transportation (DOT) regulations for hazardous and non-hazardous pharmaceutical waste.
- Disposition of the investigational product must be witnessed by two members of the research team and documented per institutional policy
- Documentation of IDS accountability will be performed from the time of initial product receipt through the destruction or return of the product to the supplier

The investigator is responsible for keeping accurate records of the clinical supplies received from Merck or designee, the amount dispensed to and returned by the participants and the amount remaining at the conclusion of the trial.

Upon completion or termination of the study, all unused and/or partially used investigational product will be destroyed at the site per institutional policy. It is the Investigator's responsibility to arrange for disposal of all empty containers, provided that procedures for proper disposal have been established according to applicable federal, state, local and institutional guidelines and procedures, and provided that appropriate records of disposal are kept.

#### 9.0 ADMINISTRATIVE AND REGULATORY DETAILS

#### 9.0.1 Confidentiality of Data

Both the investigator and the Sponsor affirm that information regarding this trial will be maintained in confidence, and such information will be divulged to the institutional review board, ethics review committee (IRB) or similar or expert committee; affiliated institution and employees, only under an appropriate understanding of confidentiality with such board or committee, affiliated institution and employees. Data generated by this trial will be considered confidential by the Sponsor and the investigator.

## 9.0.2 Confidentiality of Subject Records

The investigator agrees that the IRB or regulatory authority representatives may consult and/or copy trial documents in order to verify worksheet/case report form data. By signing the consent form, the subject agrees to this process. If trial documents will be photocopied during the process of verifying worksheet/case report form information, the subject will be identified by unique code only; full names/initials will be masked prior to transmission to the Sponsor.

The investigator and Sponsor agree to treat all subject data used and disclosed in connection with this trial in accordance with all applicable privacy laws, rules and regulations.

## 9.0.3 Confidentiality of Investigator Information

The investigator recognizes that certain personal identifying information with respect to the investigator, and all sub-investigators and trial site personnel, may be used and disclosed for trial management purposes, as part of a regulatory submission, and as required by law. This information may include:

- 1. Name, address, telephone number and e-mail address;
- 2. Hospital or clinic address and telephone number;
- 3. Curriculum vitae or other summary of qualifications and credentials; and
- 4. Other professional documentation.

Consistent with the purposes described above, this information may be transmitted to the Sponsor, and subsidiaries, affiliates and agents of the Sponsor, in your country and other countries, including countries that do not have laws protecting such information. Additionally, the investigator's name and business contact information may be included when reporting certain serious adverse events to regulatory authorities or to other investigators. By signing this protocol, the investigator expressly consents to these uses and disclosures.

# 9.0.4 Confidentiality of IRB Information

The Sponsor is required to record the name and address of each IRB that reviews and approves this trial. The Sponsor is also required to document that each IRB meets regulatory and ICH GCP requirements by requesting and maintaining records of the names and qualifications of the IRB members and to make these records available for regulatory agency review upon request by those agencies.

## 10.1 Compliance with Financial Disclosure Requirements

Financial Disclosure requirements are outlined in the US Food and Drug Administration Regulations, Financial Disclosure by Clinical Investigators (21 CFR Part 54). It is the Sponsor's responsibility to determine, based on these regulations, whether a request for Financial Disclosure information is required. It is the investigator's/subinvestigator's responsibility to comply with any such request.

The investigator/subinvestigator(s) agree, if requested by the Sponsor in accordance with 21 CFR Part 54, to provide his/her financial interests in and/or arrangements with the Sponsor to allow for the submission of complete and accurate certification and disclosure statements. The investigator/subinvestigator(s) further agree to provide this information on a Certification/Disclosure Form, commonly known as a financial disclosure form, provided by the Sponsor. The investigator/subinvestigator(s) also consent to the transmission of this information to the Sponsor in the United States for these purposes. This may involve the transmission of information to countries that do not have laws protecting personal data.

#### 10.2 Compliance with Law, Audit and Debarment

The investigator agrees to conduct the trial in an efficient and diligent manner and in conformance with this protocol; generally accepted standards of Good Clinical Practice (e.g., International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use Good Clinical Practice: Consolidated Guideline and other generally accepted standards of good clinical practice); and all applicable federal, state and local laws, rules and regulations relating to the conduct of the clinical trial.

The investigator also agrees to allow monitoring, audits, IRB review and regulatory authority inspection of trial-related documents and procedures and provide for direct access to all trial-related source data and documents.

The investigator agrees not to seek reimbursement from subjects, their insurance providers or from government programs for procedures included as part of the trial reimbursed to the investigator by the Sponsor.

The investigator shall prepare and maintain complete and accurate trial documentation in compliance with Good Clinical Practice standards and applicable federal, state and local laws, rules and regulations; and, for each subject participating in the trial, provide all data, and, upon completion or termination of the clinical trial, submit any other reports to the Sponsor as required by this protocol or as otherwise required pursuant to any agreement with the Sponsor.

Trial documentation will be promptly and fully disclosed to the Sponsor by the investigator upon request and also shall be made available at the trial site upon request for inspection, copying, review and audit at reasonable times by representatives of the Sponsor or any regulatory authorities. The investigator agrees to promptly take any reasonable steps that are requested by the Sponsor as a result of an audit to cure deficiencies in the trial documentation and worksheets/case report forms.

The investigator must maintain copies of all documentation and records relating to the conduct of the trial in compliance with all applicable legal and regulatory requirements. This documentation includes, but is not limited to, the protocol, worksheets/case report forms, advertising for subject participation, adverse

event reports, subject source data, correspondence with regulatory authorities and IRBs/ERCs, consent forms, investigator's curricula vitae, monitor visit logs, laboratory reference ranges, laboratory certification or quality control procedures and laboratory director curriculum vitae. The investigator agrees that documentation shall be retained until at least 2 years after the last approval of a marketing application in an ICH region or until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product.

Because the clinical development and marketing application process is variable, it is anticipated that the retention period can be up to 15 years or longer after protocol database lock. The Sponsor will determine the minimum retention period and notify the investigator when documents may be destroyed. The Sponsor will determine the minimum retention period and upon request, will provide guidance to the investigator when documents no longer need to be retained. The sponsor also recognizes that documents may need to be retained for a longer period if required by local regulatory requirements. All trial documents shall be made available if required by relevant regulatory authorities. The investigator must consult with and obtain written approval by the Sponsor prior to destroying trial and/or subject files.

ICH Good Clinical Practice guidelines recommend that the investigator inform the subject's primary physician about the subject's participation in the trial if the subject has a primary physician and if the subject agrees to the primary physician being informed.

The investigator will promptly inform the Sponsor of any regulatory authority inspection conducted for this trial.

Persons debarred from conducting or working on clinical trials by any court or regulatory authority will not be allowed to conduct or work on this Sponsor's trials. The investigator will immediately disclose in writing to the Sponsor if any person who is involved in conducting the trial is debarred or if any proceeding for debarment is pending or, to the best of the investigator's knowledge, threatened.

In the event the Sponsor prematurely terminates a particular trial site, the Sponsor will promptly notify that trial site's IRB.

## 11.0 Compliance with Trial Registration and Results Posting Requirements

Under the terms of the Food and Drug Administration Modernization Act (FDAMA) and the Food and Drug Administration Amendments Act (FDAAA), the Sponsor of the trial is solely responsible for determining whether the trial and its results are subject to the requirements for submission to the Clinical Trials Data Bank, http://www.clinicaltrials.gov. Information posted will allow subjects to identify potentially appropriate trials for their disease conditions and pursue participation by calling a central contact number for further information on appropriate trial locations and trial site contact information.

The Sponsor agrees to be responsible for implementing and maintaining a quality management system with written development procedures and functional area standard operating procedures (SOPs) to ensure that trials are conducted and data are generated, documented, and reported in compliance with the protocol, accepted standards of Good Clinical Practice, and all applicable federal, state, and local laws, rules and regulations relating to the conduct of the clinical trial.

The Quality Assurance (QA) division in the Miami Cancer Institute Office of Clinical Research (MCI OCR) is responsible for ensuring that industry standards of quality are met and exceeded on an on-going basis. The division is responsible for the identification, management, and prevention of quality issues, reviewing subject research charts, and mapping out current processes. They develop and implement quality and verification checks, including necessary assessment tools and checklists used during the QC process. Moreover, they facilitate and advice on corrections and corrective and preventive actions related to quality issues, provide guidance on interpretation and application of regulations, manage FDA and sponsor site visits, and work with site manager to create, implement, and evaluate action plans.

#### 12.0 DATA MANAGEMENT

The Miami Cancer Institute Office of Clinical Research (MCI OCR) oversees record keeping and handling of data is to record, store, transfer and, where necessary, convert efficiently and accurately, the information gathered on each trial subject into data.

All steps involved in data management should be documented in order to allow step-by-step retrospective assessment of quality of the data and the performance of the clinical trial (the "audit paper trail" concept). Documentation is facilitated by methods such as the use of checklists and forms giving details of action taken, dates, the individuals responsible, etc.

In the event of electronic data handling, confidentiality of the database must be secured by safety procedures such as passwords and written assurances from all staff involved. Provision must be made for the satisfactory maintenance of the database and for back-up procedures.

# 12.1 Responsibilities of the investigator

- a) The investigator has overall responsibility for ensuring the accuracy and completeness of the investigator must ensure that the observations and findings are recorded correctly and completely in the case-report forms (CRFs) and signed by the responsible person designated in the protocol. When conducting a study and using CRFs to report clinical trial data to the sponsor, the investigator must also ensure that the routine requirements for recording of data in the source documents (e.g. hospital and laboratory records, consultation files) are met, particularly those relating to the treatment given to the subject and adverse events.
- b) If trial data are entered directly into a computer, there must always be an adequate safeguard to ensure validation, including a signed and dated print-out and back-up records. Computerized systems should be validated and a detailed description for their use be produced and kept up-to-date.
- c) All corrections to CRFs and to raw data must be made in a way which does not obscure the original entry. The correct data must be inserted with the reason for the correction (if not obvious), the date, and the initials of the investigator or authorized person. For electronic data processing, only authorized persons should be permitted to enter or modify data in the computer and there should be a record of changes and deletions. If data are altered during processing, the alteration must be documented.
- d) Laboratory values with normal reference ranges, preferably together with the specificity and sensitivity of the methods used, should always be recorded on the CRF or be attached to it. Values outside a clinically accepted reference range or values that differ significantly from previous values must be evaluated and commented upon by the investigator.

- e) Data other than those required by the protocol may appear on the CRF, provided they are clearly marked as additional or optional findings, with an explanation of their significance.
- f) Units of measurement must always be stated, and conversion of units must always be stated and documented.
- g) The final report of the trial should be drawn up as defined in the protocol. The report should be signed by the sponsor, monitor and investigator(s) as well as the responsible statistician, in accordance with the applicable regulations.
- h) For a period of time defined by national regulations, the investigator should maintain a confidential record to allow the translation of the unambiguous code used to conceal the identity of the individual subjects in the trial (subject identification code). The investigator may submit the subject identification code list to the drug regulatory authority after the trial, together with the final report, according to national regulations.
- i) The investigator should ensure that the subject's participation in the clinical trial is clearly marked in his or her medical records.

#### 13.0 REFERENCES

- 1. Chung H, Ros W, Delord JP, Perets R, Italiano A, Shapira-Frommer R, et al. Efficacy and safety of pembrolizumab in previously treated advanced cervical cancer: results from the phase II Keynote- 158 study. J Clin Oncol 2019;37: 1470-1478.
- 2. Barber LJ, Sandhu S, Chen L, Campbell J, Kozarewa I, Fenwick K, et al. Secondary mutations in BRCA2 associated with clinical resistance to a PARP inhibitor. J Pathol 2013; 229(3):422-429.
- 3. Swisher EM, Sakai W, Karlan BY, Wurz K, Urban N, Taniguchi T. Secondary BRCA1 mutations in BRCA1-mutated ovarian carcinomas with platinum resistance. Cancer Res 2008; 68(8):2581-2586.
- 4. Bouwman P, Aly A, Escandell JM, Pieterse M, Bartkova J, van der Gulden H, et al. 53BP1 loss rescues BRCA1 deficiency and is associated with triple-negative and BRCA-mutated breast cancers. Nat Struct Mol Biol 2010; 17(6):688-695.
- 5. Robson M, Goessi C, Domchek S. Olaparib for Metastatic Breast Cancer in Patients with a Germline BRCA Mutation. N Engl J Med 2017;377(6):523-533.
- 6. Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, et al. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol 2017;18(3):e143-e152.
- 7. Pujade-Lauraine E, Ledermann JA, Selle F, Gebski V, Penson RT, Oza AM, et al. Olaparib tablets as maintenance therapy in patients withplatinum-sensitive, relapsed ovarian cancer and a BRCA1/2 mutation (SOLO2/ENGOTOv21):a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol 2017;18(9): 1274-1284.
- 8. Ledermann J, Pujade-Lauraine E. Olaparib maintenance therapy in platinum-sensitive relapsed ovarian cancer. N Engl J Med 2012;366(15):1382-92.

- 9. Moore KN, DiSilvestro P, Lowe ES, Garnett S, Pujade-Lauraine E SOLO1 and SOLO2: Randomized phase III trials of olaparib in patients (pts) with ovarian cancer and a BRCA1/2 mutation (BRCAm). ASCO. 2014. Chicago, IL.
- 10.Common Terminology Criteria for Adverse Events <a href="https://ctep.cancer.gov/protocoldevelopment/electronic">https://ctep.cancer.gov/protocoldevelopment/electronic</a> applications/docs/CTCAE v5 Quick Reference 8.5x11.pdf. [Accessed September 30, 2018].
- 11. Bryant HE, Schultz N, Thomas, HD, Parker KM, Flower D, Lopez E, et al. Specific killing of BRCA2-deficient tumours with inhibitors of poly (ADP-ribose) polymerase. Nature 2005;434(7035):913-7.
- 12. Farmer H, McCabe N, Lord CJ, Tutt AN, Johnson DA, Richardson TB, et al. Targeting the DNA repair defect in BRCA mutant cells as a therapeutic strategy. Nature 2005;434(7035):917-21.
- 13. Tutt A, Robson M, Garber J, Domchek S, Audeh MW, Weitzel JN, et al. Phase II trial of the oral PARP inhibitor olaparib in BRCA-deficient advanced breast cancer. J Clin Oncol 27:18s, 2009 (suppl; abstr CRA501).
- 14. Fong P, Boss D, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, et al. Inhibition of poly(ADP-ribose) polymerase in tumors from BRCA mutation carriers. N Engl J Med 2009;361(2):123-34.
- 15. Audeh MW, Carmichael J, Penson RT, Friedlander M, Powell B, Bell-McGuinn KM, et al. Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with BRCA1 or BRCA2 mutations and recurrent ovarian cancer: a proof-of-concept trial. Lancet 2010;376(9737):245-51.
- 16. Bagby GC Jr. Genetic basis of Fanconi anemia. Curr Opin Hematol 2003;10(1):68-76.
- 17. D'Andrea AD, Grompe M. The Fanconi anaemia/BRCA pathway. Nat Rev Cancer 2003;3:23-34.
- 18. Reid S, Schindler D, Hanenberg H, Barker K, Hanks S, Kalb R, et al. Biallelic mutations in PALB2 cause Fanconi anemia subtype FA-N and predispose to childhood cancer. Nat Genet 2007;39(2):162-4.
- 19. Xia B, Dorsman JC, Ameziane N, de Vries Y, Rooimans MA, Sheng Q, et al. Fanconi anemia is associated with a defect in the BRCA2 partner PALB2. Nat Genet 2007;39(2):159-61.
- 20. Smogorzewska A, Matsuoka S, Vinciguerra P, McDonald ER 3rd, Hurov KE, Luo J, et al. Identification of the FANCI protein, a monoubiquitinated FANCD2 paralog required for DNA repair. Cell 2007;129(2):289-301.
- 21. Kim Y, Lach FP, Desetty R, Hanenberg H, Auerbach AD, Smogorzewska A. Mutations of the SLX4 gene in Fanconi anemia. Nat Genet 2011; 43:138-141.
- 22. Vaz F, Hanenberg H, Schuster B, Barker K, Wiek C, Erven V, et al. Mutation of the RAD51C gene in a Fanconi anemia-like disorder. Nat Genet 2010;42:406-409.
- 23. Machida YJ, Machida Y, Chen Y, Gurtan AM, Kupfer GM, D'Andrea AD, et al. UBE2T is the E2 in the Fanconi anemia pathway and undergoes negative autoregulation. Mol Cel 2006;23(4):589-96.

- 24. Meetei AR, Yan Z, Wang W. FANCL replaces BRCA1 as the likely ubiquitin ligase responsible for FANCD2 monoubiquitination. Cell Cycle 2004;3(2):179-81.
- 25. Garcia-Higuera I, Taniguchi T, Ganesan S, Meyn MS, Timmers C, Hejna J, et al. Interaction of the Fanconi anemia proteins and BRCA1 in a common pathway. Mol Cell 2000;7(2):249-62.
- 26. Duan W, Gao L, Zhao W, Leon M, Sadee W, Webb A, et al. Assessment of FANCD2 nuclear foci formation in paraffin embedded tumors: a potential patient enrichment strategy for treatment with DNA interstrand crosslink agents. Transl Res 2013; 161(3):156-64.
- 27. Villalona-Calero MA, Duan W, Zhao W, Shilo K, Schaaf LJ, Thurmond J, et al. Veliparib Alone or in Combination with Mitomycin C in Patients with Solid Tumors With Functional Deficiency in Homologous Recombination Repair. J Natl Cancer Inst 2016;4;108(7).
- 28. Murai J, Huang SY, Das BB, Renaud A, Zhang Y, Doroshow JH, et al. Trapping of PARP1 and PARP2 by Clinical PARP Inhibitors. Cancer Res 2012; 72(21):5588-5599.
- 29. Murai J, Huang SY, Renaud A, Zhang Y, Ji J, Takeda S, et al. Stereospecific PARP trapping by BMN 673 and comparison with olaparib and rucaparib. Mol Cancer Ther 2014; 13(2):433-443.
- 30. Rottenberg S, Jaspers JE, Kersbergen A, van der Burg E, Nygren AO, Zander SA, et al. High sensitivity of *BRCA1*-deficient mammary tumors to the PARP inhibitor AZD2281 alone and in combination with platinum drugs. Proc Natl Acad Sci 2008;105(44):17079-84.
- 31. Hay T, Matthews JR, Pietzka L, Lau A, Cranston A, Nygren AO, et al. Poly(ADP-ribose) polymerase-1 inhibitor treatment regresses autochthonous Brca2/p53-mutant mammary tumors in vivo and delays tumor relapse in combination with carboplatin. Cancer Res 2009;69(9):3850-5.
- 32. Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, et al. Inhibition of poly(ADP-ribose) polymerase in tumors from *BRCA* mutation carriers. N Engl J Med 2009;361(2):123-34.
- 33. Helleday T. The underlying mechanism for the PARP and *BRCA* synthetic lethality: Clearing up the misunderstandings. Mol Oncol 2011; 5: 387-393.
- 34. Disis ML. Immune regulation of cancer. J Clin Oncol 2010;28(29):4531-8.
- 35. Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, et al. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol 2005;23(10):2346-57.
- 36. Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, et al. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med 2008;358(25):2698-703.
- 37. Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol 2005;23:515-48.

- 38. Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A 2001;98(24):13866-71.
- 39. Zhang X, Schwartz J-CD, Guo X, Bhatia S, Cao E, Chen L, et al. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity 2004;20:337-47.
- 40. Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol 2004;173:945-54.
- 41. Sheppard K-A, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, et al. PD-1 inhibits T-cell receptor induced phosphorylation of the ZAP70/CD3zeta signalosome and downstream signaling to PKCtheta. FEBS Lett. 2004;574:37-41.
- 42. Riley JL. PD-1 signaling in primary T cells. Immunol Rev 2009;229:114-25.
- 43. Parry RV, Chemnitz JM, Frauwirth KA, Lanfranco AR, Braunstein I, Kobayashi SV, et al. CTLA-4 and PD-1 receptors inhibit T-cell activation by distinct mechanisms. Mol Cell Biol 2005;25(21):9543-53.
- 44. Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev 2010;236:219-42.
- 45. Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T. Olaparib as maintenance treatment following first-line platinum-based chemotherapy in patients with a germline BRCA mutation and metastatic pancreatic cancer: phase III POLO trial. Ann Oncol, 2019;20:152.
- 46. Le DT, Uram J, Wang H, Bartlett BC, Kemberling H, Eyring AD, et al. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20.
- 47. Vergote I, Sehouli J, Salutari V, Zola P, Madry R, Wenham RM, et al. ENGOT-OV43/KEYLYNK-001: A phase III, randomized, double-blind, active- and placebo-controlled study of pembrolizumab plus chemotherapy with olaparib maintenance for first-line treatment of BRCA-nonmutated advanced epithelial ovarian cancer. J Clin Oncol 2019 37:15 suppl), TPS5603-TPS5603.
- 48. Howlader N, Noone AM, Krapcho M, Miller D, Brest A, Yu M, et al. (eds). SEER Cancer Statistics Review, 1975-2014, National Cancer Institute, Bethesda, MD, http://seer.cancer.gov/csr/1975\_2014/, based on November 2016 SEER data submission, posted to the SEER website April 2017.
- 49. Rizvi, NA, Hellman MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, et al. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science 2015. 348(6230): 124-8.
- 50. Snyder, A. Makarov V, Merghoub T, Yuan J, Zaretsky JM, Desrichard A, et al., Genetic basis for clinical response to CTLA-4 blockade in melanoma. N Engl J Med 2014 371(23): p. 2189-2199.
- 51. Van Allen EM, Miao D, Schilling B, Shukla SA, Blank C, Zimmer L, et al., Genomic correlates of response to CTLA-4 blockade in metastatic melanoma. Science 2015;350(6257):207-211.

- 52. A'Hern, R. P. A. 2001. 'Sample size tables for exact single-stage phase II designs.' Statistics in Medicine, Volume 20, pages 859-866.
- 53. Fleming, T. R. 1982. 'One-sample multiple testing procedure for Phase II clinical trials.'Biometrics, Volume 38, pages 143-151.

## 14.0 APPENDICES

# **Appendix 1: ECOG Performance Status**

| Grade | Description |
|---|---|
| 0 | Normal activity. Fully active, able to carry on all pre-disease |
| | performance without restriction. |
| | Symptoms, but ambulatory. Restricted in physically strenuous |
| 1 | activity, but ambulatory and able to carry out work of a light or |
| | sedentary nature (e.g., light housework, office work). |
| | In bed <50% of the time. Ambulatory and capable of all self-care, but |
| 2 | unable to carry out any work activities. Up and about more than 50% |
| | of waking hours. |
| 3 | In bed >50% of the time. Capable of only limited self-care, confined |
| | to bed or chair more than 50% of waking hours. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any self-care. |
| | Totally confined to bed or chair. |
| 5 | Dead. |

<sup>\*</sup>As published in Am. J. Clin. Oncol.: Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982. The Eastern Cooperative Oncology Group, Robert Comis M.D., Group Chair.
# Appendix 2: Common Terminology Criteria for Adverse Events V5.0 (CTCAE)

The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for adverse event reporting. (http://ctep.cancer.gov/reporting/ctc.html)

For each episode of an adverse event, all changes to the CTCAE grade attained as well as the highest attained CTC grade should be reported.

# **Appendix 3: Contraceptive Guidance and Pregnancy Testing**

Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming post-menopausal unless permanently sterile (see below)

Women in the following categories are not considered WOCBP:

- Premenarchal
- Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - o Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

- Postmenopausal female
  - A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
    - A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with two FSH measurements in the postmenopausal range is required. Postmenopausal is defined as:
      - Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
      - Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50
      - radiation-induced oophorectomy with last menses >1 year ago
      - chemotherapy-induced menopause with >1 year interval since last menses
      - surgical sterilisation (bilateral oophorectomy or hysterectomy)
  - Females on HRT and whose menopausal status is in doubt will be required to use one of the non-hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

## **Contraception Requirements**

# **Female Participants:**

Female participants of childbearing potential are eligible to participate if they agree to use a highly effective method of contraception that has a low user dependency consistently and correctly as described in Table 9 during the protocol-defined time frame.

# **Acceptable Birth Control Methods**

# Olaparib is regarded as a compound with medium/high fetal risk.

Women of childbearing potential and their partners, who are sexually active, must agree to the use of TWO highly effective forms of contraception in combination [as listed below]. This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 1 month after last dose of study drug(s), or they must totally/truly abstain from any form of sexual intercourse (see below).

# Acceptable Non-hormonal birth control methods include:

- Total/True abstinence: When the patient refrains from any form of sexual intercourse and this is in line with their usual and/or preferred lifestyle; this must continue for the total duration of the trial and for at least 1 month after the last dose of study drug. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods, or declaration of abstinence solely for the duration of a trial) and withdrawal are not acceptable methods of contraception]
- Vasectomised sexual partner PLUS male condom. With participant assurance that partner received post-vasectomy confirmation of azoospermia.
- Tubal occlusion PLUS male condom
- IUD PLUS male condom. Provided coils are copper-banded

# **Acceptable hormonal methods:**

- Normal and low dose combined oral pills PLUS male condom
- Cerazette (desogestrel) PLUS male condom. Cerazette is currently the only highly efficacious progesterone based pill.
- Hormonal shot or injection (eg., Depo-Provera) PLUS male condom
- Etonogestrel implants (e.g., Implanon, Norplant) PLUS male condom
- Norelgestromin / EE transdermal system PLUS male condom
- Intrauterine system [IUS] device (eg., levonorgestrel releasing IUS -Mirena®) PLUS male condom Intravaginal device (e.g., EE and etonogestrel) PLUS male condom

# Table 16 Highly-Effective Contraceptive Methods That Have Low User Dependency

## **Highly Effective Methods That Have Low User Dependency**

Failure rate of <1% per year when used consistently and correctly.

- Progestogen- only contraceptive implant a, b
- Intrauterine hormone-releasing system (IUS) b
- Intrauterine device (IUD)
- Bilateral tubal occlusion

#### • Vasectomized partner

A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

#### • Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

#### Notes:

Use should be consistent with local regulations regarding the use of contraceptive methods for participants of clinical studies.

- a) If locally required, in accordance with Clinical Trial Facilitation Group (CTFG) guidelines, acceptable contraceptive implants are limited to those which inhibit ovulation.
- b) If hormonal contraception efficacy is potentially decreased due to interaction with study treatment, condoms must be used in addition to the hormonal contraception during the treatment period and for at least [X days, corresponding to time needed to eliminate study treatment plus 30 days for study treatments with genotoxic potential] after the last dose of study treatment.

# **Pregnancy Testing**

WOCBP should only be included after a negative highly sensitive urine or serum pregnancy test.

Pregnancy testing will be performed whenever an expected menstrual cycle is missed or when pregnancy is otherwise suspected.

# Appendix 4: Description of the iRECIST Process for Assessment of Disease Progression

Assessment at Screening and Prior to RECIST 1.1 Progression

Until radiographic progression based on RECIST 1.1, there is no distinct iRECIST assessment.

Assessment and Decision at RECIST 1.1 Progression

In participants who show evidence of radiological PD by RECIST 1.1 the Investigator will decide whether to continue a participant on study treatment until repeat imaging is obtained (using iRECIST for participant management (see Table 5 and Figures 1 and 3). This decision by the Investigator should be based on the participant's overall clinical condition.

Clinical stability is defined as the following:

- Absence of symptoms and signs indicating clinically significant progression of disease
- No decline in ECOG performance status
- No requirements for intensified management, including increased analgesia, radiation, or other palliative care

Any participant deemed clinically unstable should be discontinued from study treatment at site-assessed first radiologic evidence of PD and is not required to have repeat tumor imaging for confirmation of PD by iRECIST.

If the Investigator decides to continue treatment, the participant may continue to receive study treatment and the tumor assessment should be repeated 4 to 8 weeks later to confirm PD by iRECIST, per Investigator assessment. I

Tumor flare may manifest as any factor causing radiographic progression per RECIST 1.1, including:

- Increase in the sum of diameters of target lesion(s) identified at baseline to  $\geq 20\%$  and  $\geq 5$  mm from nadir
  - Please note: the iRECIST publication uses the terminology "sum of measurements", but "sum of diameters" will be used in this protocol, consistent with the original RECIST 1.1 terminology.
- Unequivocal progression of non-target lesion(s) identified at baseline
- Development of new lesion(s)

iRECIST defines new response categories, including iUPD (unconfirmed progressive disease) and iCPD (confirmed progressive disease). For purposes of iRECIST assessment, the first visit showing progression according to RECIST 1.1 will be assigned a visit (overall) response of iUPD, regardless of which factors caused the progression.

At this visit, target and non-target lesions identified at baseline by RECIST 1.1 will be assessed as usual.

New lesions will be classified as measurable or non-measurable, using the same size thresholds and rules as for baseline lesion assessment in RECIST 1.1. From measurable new lesions, up to 5 lesions total (up to 2 per organ), may be selected as New Lesions – Target. The sum of diameters of these lesions will be calculated and kept distinct from the sum of diameters for target lesions at baseline. All other new lesions will be followed qualitatively as New Lesions – Non-target.

# Assessment at the Confirmatory Imaging

On the confirmatory imaging, the participant will be classified as progression confirmed (with an overall response of iCPD), or as showing persistent unconfirmed progression (with an overall response of iUPD), or as showing disease stability or response (iSD/iPR/iCR).

# Confirmation of Progression

Progression is considered confirmed, and the overall response will be iCPD, if ANY of the following occurs:

- Any of the factors that were the basis for the initial iUPD show worsening
  - $\circ$  For target lesions, worsening is a further increase in the sum of diameters of  $\geq 5$  mm, compared to any prior iUPD time point
  - o For non-target lesions, worsening is any significant growth in lesions overall, compared to a prior iUPD time point; this does not have to meet the "unequivocal" standard of RECIST 1.1
  - o For new lesions, worsening is any of these:
    - An increase in the new lesion sum of diameters by  $\geq 5$  mm from a prior iUPD time point
    - Visible growth of new non-target lesions
    - The appearance of additional new lesions
- Any new factor appears that would have triggered PD by RECIST 1.1

#### Persistent iUPD

Progression is considered not confirmed, and the overall response remains iUPD, if:

- None of the progression-confirming factors identified above occurs AND
- The target lesion sum of diameters (initial target lesions) remains above the initial PD threshold (by RECIST 1.1)

Additional imaging for confirmation should be scheduled 4 to 8 weeks from the scan on which iUPD is seen. This may correspond to the next visit in the original visit schedule. The assessment of the subsequent confirmation scan proceeds in an identical manner, with possible outcomes of iCPD, iUPD, and iSD/iPR/iCR.

#### Resolution of iUPD

Progression is considered not confirmed, and the overall response becomes iSD/iPR/iCR, if:

- None of the progression-confirming factors identified above occurs, AND
- The target lesion sum of diameters (initial target lesions) is not above the initial PD threshold.

The response is classified as iSD or iPR (depending on the sum of diameters of the target lesions), or iCR if all lesions resolve.

In this case, the initial iUPD is considered to be pseudo-progression, and the level of suspicion for progression is "reset". This means that the next visit that shows radiographic progression, whenever it occurs, is again classified as iUPD by iRECIST, and the confirmation process is repeated before a response of iCPD can be assigned.

Management Following the Confirmatory Imaging

If repeat imaging does not confirm PD per iRECIST, as assessed by the Investigator, and the participant continues to be clinically stable, study treatment may continue and follow the regular imaging schedule. If PD is confirmed, participants will be discontinued from study treatment.

NOTE: If a participant has confirmed radiographic progression (iCPD) as defined above, but the participant is achieving a clinically meaningful benefit, an exception to continue study treatment may be considered. In this case, if study treatment is continued, tumor imaging should continue to be performed following the intervals as outlined in Section 6.

Detection of Progression at Visits After Pseudo-progression Resolves

After resolution of pseudo-progression (ie, achievement of iSD/iPR/iCR), iUPD is indicated by any of the following events:

- Target lesions
  - Sum of diameters reaches the PD threshold (≥ 20% and ≥ 5 mm increase from nadir) either for the first time, or after resolution of previous pseudo-progression. The nadir is always the smallest sum of diameters seen during the entire trial, either before or after an instance of pseudo-progression.
- Non-target lesions
  - o If non-target lesions have never shown unequivocal progression, their doing so for the first time results in iUPD.
  - o If non-target lesions had shown previous unequivocal progression, and this progression has not resolved, iUPD results from any significant further growth of non-target lesions, taken as a whole.
- New lesions
  - o New lesions appear for the first time
  - o Additional new lesions appear
  - $\circ$  Previously identified new target lesions show an increase of  $\geq 5$  mm in the new lesion sum of diameters, from the nadir value of that sum

o Previously identified non-target lesions show any significant growth

If any of the events above occur, the overall response for that visit is iUPD, and the iUPD evaluation process (see Assessment at the Confirmatory Imaging above) is repeated. Progression must be confirmed before iCPD can occur.

The decision process is identical to the iUPD confirmation process for the initial PD, except in one respect. If new lesions occurred at a prior instance of iUPD, and at the confirmatory scan the burden of new lesions has increased from its smallest value (for new target lesions, their sum of diameters is  $\geq 5$  mm increased from its nadir), then iUPD cannot resolve to iSD or iPR. It will remain iUPD until either a decrease in the new lesion burden allows resolution to iSD or iPR, or until a confirmatory factor causes iCPD.

Additional details about iRECIST are provided in the iRECIST publication [Seymour et al., 2017].

# Appendix 5: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### 14.1.1 Definition of AE

#### AE definition

- An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
- NOTE: For purposes of AE definition, study intervention (also referred to as Merck product) includes any pharmaceutical product, biological product, vaccine, diagnostic agent, or protocol specified procedure whether investigational or marketed (including placebo, active comparator product, or run-in intervention), manufactured by, licensed by, provided by, or distributed by Merck for human use in this study.

# **Events meeting the AE definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g., ECG, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator.
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication.
- For all reports of overdose (whether accidental or intentional) with an associated AE, the AE term should reflect the clinical symptoms or abnormal test result. An overdose without any associated clinical symptoms or abnormal laboratory results is reported using the terminology "accidental or intentional overdose without adverse effect."

## **Events NOT meeting the AE definition**

- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.
- Surgery planned prior to informed consent to treat a pre-existing condition that has not worsened.

#### 14.1.2 Definition of SAE

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met.

# An SAE is defined as any untoward medical occurrence that, at any dose:

#### a. Results in death

## b. Is life-threatening

The term "life-threatening" in the definition of "serious" refers to an event in which the participant
was at risk of death at the time of the event. It does not refer to an event, which hypothetically
might have caused death, if it were more severe.

# c. Requires inpatient hospitalization or prolongation of existing hospitalization

Hospitalization is defined as an inpatient admission, regardless of length of stay, even if the
hospitalization is a precautionary measure for continued observation. (Note: Hospitalization for an
elective procedure to treat a pre-existing condition that has not worsened is not an SAE. A preexisting condition is a clinical condition that is diagnosed prior to the use of a Merck product and
is documented in the participant's medical history.

# d. Results in persistent or significant disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (eg, sprained ankle) that may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### e. Is a congenital anomaly/birth defect

• In offspring of participant taking the product regardless of time to diagnosis.

# f. Other important medical events

- Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately lifethreatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent 1 of the other outcomes listed in the above definition. These events should usually be considered serious.
- Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

## 14.1.3 Additional Events Reported in the Same Manner as SAE

## Additional events that require reporting in the same manner as SAE

In addition to the above criteria, AEs meeting either of the below criteria, although not serious per ICH definition, are reportable to Merck in the same time frame as SAEs to meet certain local requirements. Therefore, these events are considered serious by Merck for collection purposes.

- Is a new cancer (that is not a condition of the study)
- Is associated with an overdose of pembrolizumab

## 14.1.4 Recording AE and SAE

# AE and SAE recording

- When an AE/SAE occurs, it is the responsibility of the investigator to review all documentation (eg, hospital progress notes, laboratory, and diagnostics reports) related to the event.
- The investigator will record all relevant AE/SAE information on the AE CRFs/worksheets at each examination.
- There may be instances when copies of medical records for certain cases are requested by the Merck. In this case, all participant identifiers, with the exception of the participant number, will be blinded on the copies of the medical records before submission to the Merck.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or
  other clinical information. In such cases, the diagnosis (not the individual signs/symptoms) will be
  documented as the AE/SAE.

#### Assessment of intensity/toxicity

• An event is defined as "serious" when it meets at least 1 of the predefined outcomes as described in the definition of an SAE, not when it is rated as severe.

- 1. The investigator will make an assessment of intensity for each AE and SAE (and other reportable safety event) according to the NCI Common Terminology for Adverse Events (CTCAE), version 5. Any AE that changes CTCAE grade over the course of a given episode will have each change of grade recorded on the AE CRFs/worksheets.
  - Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  - Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL).
  - Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL.
  - Grade 4: Life threatening consequences; urgent intervention indicated.
  - Grade 5: Death related to AE.

# **Assessment of causality**

- 1. Did Merck product cause the AE?
- 2. The determination of the likelihood that Merck product caused the AE will be provided by an investigator who is a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test product and the AE based upon the available information.
- 3. The following components are to be used to assess the relationship between Merck's product and the AE; the greater the correlation with the components and their respective elements (in number and/or intensity), the more likely Merck product caused the AE:
  - Exposure: Is there evidence that the participant was actually exposed to Merck product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen?
  - **Time Course:** Did the AE follow in a reasonable temporal sequence from administration of Merck product? Is the time of onset of the AE compatible with a drug-induced effect (applies to studies with investigational medicinal product)?
  - **Likely Cause:** Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s)/vaccine(s), or other host or environmental factors.
  - **Dechallenge:** Was Merck product discontinued or dose/exposure/frequency reduced?
  - If yes, did the AE resolve or improve?
  - If yes, this is a positive dechallenge.

- If no, this is a negative dechallenge.
- (Note: This criterion is not applicable if: (1) the AE resulted in death or permanent disability; (2) the AE resolved/improved despite continuation of the Merck product; (3) the study is a single-dose drug study; or (4) Merck product(s) is/are only used 1 time.)
- **Rechallenge:** Was the participant re-exposed to Merck product in this study?
- If yes, did the AE recur or worsen?
- If yes, this is a positive rechallenge.
- If no, this is a negative rechallenge.

(Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) the study is a single-dose drug study; or (3) Merck product(s) is/are used only 1 time.)

NOTE: IF A RECHALLENGE IS PLANNED FOR AN AE THAT WAS SERIOUS AND MAY HAVE BEEN CAUSED BY MERCK PRODUCT, OR IF RE-EXPOSURE TO MERCK'S PRODUCT POSES ADDITIONAL POTENTIAL SIGNIFICANT RISK TO THE PARTICIPANT THEN THE RECHALLENGE MUST BE APPROVED IN ADVANCE BY THE SPONSOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL, AND IF REQUIRED, THE INIRB/IEC.

- 4. **Consistency with study intervention profile:** Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding Merck product or drug class pharmacology or toxicology?
- 5. The assessment of relationship will be reported on the case report forms/worksheets by an investigator who is a qualified physician according to his/her best clinical judgment, including consideration of the above elements.
- 6. Use the following scale of criteria as guidance (not all criteria must be present to be indicative of Merck product relationship).
  - Yes, there is a reasonable possibility of Merck product relationship:
  - There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the administration of Merck product is reasonable. The AE is more likely explained by Merck product than by another cause.
  - No, there is not a reasonable possibility of Merck product relationship:
  - Participant did not receive the Merck product OR temporal sequence of the AE onset relative to administration of the Merck product is not reasonable OR the AE is more likely explained by another cause than the Merck product. (Also entered for a participant with overdose without an associated AE.)

- 7. For each AE/SAE, the investigator must document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- 8. There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the Merck. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to Merck.
- 9. The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- 10. The causality assessment is 1 of the criteria used when determining regulatory reporting requirements.
- 11. For studies in which multiple agents are administered as part of a combination regimen, the investigator may attribute each AE causality to the combination regimen or to a single agent of the combination. In general, causality attribution should be assigned to the combination regimen (ie, to all agents in the regimen). However, causality attribution may be assigned to a single agent if, in the investigator's opinion, there is sufficient data to support full attribution of the AE to the single agent.

# Follow-up of AE and SAE

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.
- New or updated information will be recorded in the CRF.
- The investigator will submit any updated SAE data to Merck within 2 business days but no longer than 3 calendar days of receipt of the information.

# 14.1.5 Reporting of AEs, SAEs, and Other Reportable Safety Events to the Merck

SAE reports and any other relevant safety information are to be forwarded to the Merck Global Safety facsimile number: +1-215-661-6229

A copy of all 15 Day Reports and Annual Progress Reports is submitted as required by FDA, European Union (EU), Pharmaceutical and Medical Devices agency (PMDA) or other local regulators. Investigators will cross-reference this submission according to local regulations to the Merck Investigational Compound Number (IND, CSA, etc.) at the time of submission. Additionally, investigators will submit a copy of these reports to Merck & Co., Inc. (Attn: Worldwide Product Safety; FAX 215-661-6229) at the time of submission to FDA.